CLINICAL TRIAL: NCT04857892
Title: A Two-Part, Randomized, Open-Label, Single Dose, Crossover Clinical Study to Assess the Relative Bioavailability of Fixed-Dose Combinations of GSK3640254 and Dolutegravir and to Assess the Effect of Food on the Select Fixed Dose Combination of GSK3640254 and Dolutegravir in Healthy Participants
Brief Title: A Relative Bioavailability and Food-Effect Study of the Fixed Dose Combination of GSK3640254 and Dolutegravir (DTG) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 213055
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-08

CONDITIONS: HIV Infections
Keywords: Dolutegravir; GSK3640254; Fixed Dose Combinations; Bioavailability
MeSH Terms: conditions — HIV Infections | interventions — GSK3640254

STUDY DESIGN:
Intervention Model Description: This is a 2-part crossover study.
Masking Description: This is an open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1 : Treatment sequence ABC (Experimental): Participants will receive a single oral dose of GSK3640254 25 milligrams (mg) (2 x tablets), GSK3640254 100 mg (1 x tablet) and DTG 50 mg (1 x tablet) administered together under moderate fat and calorie conditions (reference) (Treatment A) in Period 1, followed by a single oral dose of GSK3640254/DTG, 150 mg/50 mg (1 x monolayer tablet) FDC administered under moderate fat and calorie conditions (Treatment B) in Period 2. In Period 3, participants will receive a single oral dose of GSK3640254 / DTG, 150 mg/50 mg (1 x bilayer tablet) FDC administered under moderate fat and calorie conditions (Treatment C).
  Interventions: Drug: GSK3640254; Drug: DTG; Drug: GSK3640254/DTG
- Part 1 : Treatment sequence BCA (Experimental): Participants will receive a single oral dose of GSK3640254/DTG, 150 mg/50 mg (1 x monolayer tablet) FDC administered under moderate fat and calorie conditions (Treatment B) in Period 1, followed by a single oral dose of GSK3640254 / DTG, 150 mg/50 mg (1 x bilayer tablet) FDC administered under moderate fat and calorie conditions (Treatment C) in Period 2. In Period 3 participants will receive a single oral dose of GSK3640254 25 mg (2 x tablets), GSK3640254 100 mg (1 x tablet) and DTG 50 mg (1 x tablet) administered together under moderate fat and calorie conditions (reference) (Treatment A).
  Interventions: Drug: GSK3640254; Drug: DTG; Drug: GSK3640254/DTG
- Part 1 : Treatment sequence CAB (Experimental): Participants will receive a single oral dose of GSK3640254 / DTG, 150 mg/50 mg (1 x bilayer tablet) FDC administered under moderate fat and calorie conditions (Treatment C) in period 1, followed by a single oral dose of GSK3640254 25 mg (2 x tablets), GSK3640254 100 mg (1 x tablet) and DTG 50 mg (1 x tablet) administered together under moderate fat and calorie conditions (reference) (Treatment A) in Period 2. In Period 3 participants will receive a single oral dose of GSK3640254/DTG, 150 mg/50 mg (1 x monolayer tablet) FDC administered under moderate fat and calorie conditions (Treatment B).
  Interventions: Drug: GSK3640254; Drug: DTG; Drug: GSK3640254/DTG
- Part 2 : Treatment sequence DE (Experimental): Participants will receive a single oral dose of selected FDC from Part 1 of GSK3640254/DTG, 150 mg/50 mg administered under high fat and calorie conditions (Treatment D) in Period 1 followed by a single oral dose of selected FDC from Part 1 of GSK3640254/DTG, 150 mg/50 mg administered under fasted conditions (Treatment E) in Period 2.
  Interventions: Drug: GSK3640254/DTG
- Part 2 : Treatment sequence ED (Experimental): Participants will receive a single oral dose of selected FDC from Part 1 of GSK3640254/DTG, 150 mg/50 mg administered under fasted conditions (Treatment E) in Period 1 followed by a single oral dose of selected FDC from Part 1 of GSK3640254/DTG, 150 mg/50 mg administered under high fat and calorie conditions (Treatment D) in Period 2.
  Interventions: Drug: GSK3640254/DTG

INTERVENTIONS:
Drug: GSK3640254 — GSK3640254 will be administered via oral route.
  Arms: Part 1 : Treatment sequence ABC; Part 1 : Treatment sequence BCA; Part 1 : Treatment sequence CAB
Drug: DTG — DTG will be administered via oral route.
  Arms: Part 1 : Treatment sequence ABC; Part 1 : Treatment sequence BCA; Part 1 : Treatment sequence CAB
Drug: GSK3640254/DTG — GSK3640254/DTG will be administered via oral route.

SUMMARY:
This is a two part study to compare the relative bioavailability (BA) of 2 fixed dose combinations (FDCs) of GSK3640254/DTG with GSK3640254 and DTG administered together as single agents (Part 1) and to assess the effect of food on the pharmacokinetic (PK) of the selected FDC of GSK3640254/DTG (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 65 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring (history and ECG).
* Participants capable of giving signed informed consent.

Exclusion Criteria:

* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A pre-existing condition interfering with normal gastro intestinal anatomy or motility (for example [e.g.], gastroesophageal reflux disease, gastric ulcers, gastritis) or hepatic and/or renal function that could interfere with the absorption, metabolism, and/or excretion of the study intervention or render the participant unable to take oral study intervention.
* Prior cholecystectomy surgery (prior appendectomy is acceptable).
* Clinically significant illness, including viral syndromes within 3 weeks of dosing.
* Participant with known or suspected active Coronavirus disease (COVID)-19 infection or contact with an individual with known COVID-19, within 14 days of study enrollment.
* Current enrollment or past participation within the last 30 days before signing of consent in any other clinical study involving an investigational study intervention (including an investigational COVID vaccine) or any other type of medical research.
* Prior exposure to GSK3640254 or prior intolerance to DTG in this or another clinical study.
* Any positive (abnormal) response confirmed by the investigator on a screening clinician- or qualified designee-administered Columbia Suicide Severity Rating Scale (C-SSRS).
* Any significant arrhythmia or ECG finding (e.g., prior myocardial infarction in the past 3 months, symptomatic bradycardia, non-sustained or sustained atrial arrhythmias, non-sustained or sustained ventricular tachycardia, any degree of atrioventricular block, or conduction abnormality) which, in the opinion of the investigator or ViiV Healthcare (VH)/GlaxoSmithKline (GSK) medical monitor, will interfere with the safety for the individual participant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, open-label, single dose, crossover clinical study to assess relative bioavailability and food-effect of the fixed dose combination (FDC) of GSK3640254 and Dolutegravir (DTG) in healthy participants.
Pre-assignment Details: A total of 41 participants (23 participants in Part 1 and 18 participants in Part 2) were enrolled in the study.
Groups:
- Part 1: Cohort 1: Sequence ABC: Participants received Treatment A as a single oral dose of GSK3640254 25 milligrams (mg) (2 tablets), GSK3640254 100 mg (1 tablet)/dolutegravir (DTG) 50 mg (1 tablet) administered together under moderate fat and calorie conditions on Day 1 in treatment period 1 followed by Treatment B as a single oral dose of GSK3640254/DTG, 150 mg/50 mg (1 monolayer tablet) FDC administered under moderate fat and calorie conditions on Day 1 in treatment period 2, further followed by Treatment C as a single oral dose of GSK3640254/DTG, 150 mg/50 mg (1 bilayer tablet) FDC administered under moderate fat and calorie conditions on Day 1 in treatment period 3. There was washout period of 7 days between each treatment period.
- Part 1: Cohort 2: Sequence BCA: Participants received Treatment B as a single oral dose of GSK3640254/DTG, 150 mg/50 mg (1 monolayer tablet) FDC administered under moderate fat and calorie conditions on Day 1 in treatment period 1 followed by Treatment C as a single oral dose of GSK3640254/DTG, 150 mg/50 mg (1 bilayer tablet) FDC administered under moderate fat and calorie conditions on Day 1 in treatment period 2, further followed by Treatment A as a single oral dose of GSK3640254 25 mg (2 tablets), GSK3640254 100 mg (1 tablet), and DTG 50 mg (1 tablet) administered together under moderate fat and calorie conditions on Day 1 on treatment period 3. There was washout period of 7 days between each treatment period.
- Part 1: Cohort 3: Sequence CAB: Participants received Treatment C as a single oral dose of GSK3640254/DTG, 150 mg/50 mg (1 bilayer tablet) FDC administered under moderate fat and calorie conditions on Day 1 in treatment period 1 followed by Treatment A as a single oral dose of GSK3640254 25 mg (2 tablets), GSK3640254 100 mg (1 tablet) and DTG 50 mg (1 tablet) administered together under moderate fat and calorie conditions (reference) on Day 1 in treatment period 2, further followed by Treatment B as a single oral dose of GSK3640254/DTG, 150 mg/50 mg (1 monolayer tablet) FDC administered under moderate fat and calorie conditions on Day 1 in treatment period 3. There was washout period of 7 days between each treatment period.
- Part 2: Cohort 1: Sequence DE: Participants received Treatment D as a single oral dose of selected bilayer FDC from Part 1 of GSK3640254/DTG, 150 mg/50 mg administered under high fat and calorie conditions on Day 1 in treatment Period 1, followed by Treatment E as a single oral dose of selected FDC of GSK3640254/DTG, 150 mg/50 mg administered under fasted conditions on Day 1 in treatment Period 2. There was washout period of 7 days between each treatment period.
- Part 2: Cohort 2: Sequence ED: Participants received Treatment E as a single oral dose of selected bilayer FDC from Part 1 of GSK3640254/DTG, 150 mg/50 mg administered under fasted conditions on Day 1 in treatment Period 1, followed by Treatment D as a single oral dose of selected FDC of GSK3640254/DTG, 150 mg/50 mg administered under high fat and calorie conditions on Day 1 in treatment Period 2. There was washout period of 7 days between each treatment period.
Period: Part 1: Period 1 (Day 1)
Arm/Group | Part 1: Cohort 1: Sequence ABC | Part 1: Cohort 2: Sequence BCA | Part 1: Cohort 3: Sequence CAB | Part 2: Cohort 1: Sequence DE | Part 2: Cohort 2: Sequence ED
Started | 9 | 7 | 7 | 0 | 0
Completed | 8 | 7 | 7 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Period: Part 1: Washout Period 1 (Up to 7 Days)
Arm/Group | Part 1: Cohort 1: Sequence ABC | Part 1: Cohort 2: Sequence BCA | Part 1: Cohort 3: Sequence CAB | Part 2: Cohort 1: Sequence DE | Part 2: Cohort 2: Sequence ED
Started | 8 | 7 | 7 | 0 | 0
Completed | 8 | 7 | 7 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 1: Period 2 (Day 1)
Arm/Group | Part 1: Cohort 1: Sequence ABC | Part 1: Cohort 2: Sequence BCA | Part 1: Cohort 3: Sequence CAB | Part 2: Cohort 1: Sequence DE | Part 2: Cohort 2: Sequence ED
Started | 8 | 7 | 7 | 0 | 0
Completed | 8 | 7 | 7 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 1: Washout Period 2 (Up to 7 Days)
Arm/Group | Part 1: Cohort 1: Sequence ABC | Part 1: Cohort 2: Sequence BCA | Part 1: Cohort 3: Sequence CAB | Part 2: Cohort 1: Sequence DE | Part 2: Cohort 2: Sequence ED
Started | 8 | 7 | 7 | 0 | 0
Completed | 6 | 6 | 6 | 0 | 0
Not Completed | 2 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0 | 0
Period: Part 1: Period 3 (Day 1)
Arm/Group | Part 1: Cohort 1: Sequence ABC | Part 1: Cohort 2: Sequence BCA | Part 1: Cohort 3: Sequence CAB | Part 2: Cohort 1: Sequence DE | Part 2: Cohort 2: Sequence ED
Started | 6 | 6 | 6 | 0 | 0
Completed | 6 | 6 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 2: Period 1 (Day 1)
Arm/Group | Part 1: Cohort 1: Sequence ABC | Part 1: Cohort 2: Sequence BCA | Part 1: Cohort 3: Sequence CAB | Part 2: Cohort 1: Sequence DE | Part 2: Cohort 2: Sequence ED
Started | 0 | 0 | 0 | 9 | 9
Completed | 0 | 0 | 0 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 2: Washout Period 1 (Up to 7 Days)
Arm/Group | Part 1: Cohort 1: Sequence ABC | Part 1: Cohort 2: Sequence BCA | Part 1: Cohort 3: Sequence CAB | Part 2: Cohort 1: Sequence DE | Part 2: Cohort 2: Sequence ED
Started | 0 | 0 | 0 | 9 | 9
Completed | 0 | 0 | 0 | 9 | 8
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Period: Part 2: Period 2 (Day 1)
Arm/Group | Part 1: Cohort 1: Sequence ABC | Part 1: Cohort 2: Sequence BCA | Part 1: Cohort 3: Sequence CAB | Part 2: Cohort 1: Sequence DE | Part 2: Cohort 2: Sequence ED
Started | 0 | 0 | 0 | 9 | 8
Completed | 0 | 0 | 0 | 9 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Cohort 1: Sequence ABC | Part 1: Cohort 2: Sequence BCA | Part 1: Cohort 3: Sequence CAB | Part 2: Cohort 1: Sequence DE | Part 2: Cohort 2: Sequence ED | Total
Number analyzed (Participants) | 9 | 7 | 7 | 9 | 9 | 41
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  19-64 years | 9 | 7 | 7 | 9 | 9 | 41
  >= 65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 5 | 2 | 18
  Male | 6 | 3 | 3 | 4 | 7 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 3 | 3 | 3 | 6 | 3 | 18
  White-White/Caucasian/European Heritage | 6 | 3 | 4 | 3 | 4 | 20
  Multiple | 0 | 1 | 0 | 0 | 0 | 1
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian- South East Asian Heritage | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Area Under the Plasma Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC[0-inf]) of GSK3640254
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of GSK3640254.
Time Frame: Pre-dose, 30 minutes, 1 hour, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72, 96 hours post dose in each treatment period
Population: PK Parameter Population consisted of all participants who underwent plasma PK sampling and had evaluable PK parameters estimated. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Groups:
- Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg: Participants received a single oral dose of GSK3640254 25 mg (2 tablets), GSK3640254 100 mg (1 tablet), and DTG 50 mg (1 tablet) together under moderate fat and calorie conditions on Day 1 in treatment period 1, 2 and 3.
- Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet): Participants received a single oral dose of GSK3640254 / DTG, 150 mg/50 mg (1 monolayer tablet) FDC under moderate fat and calorie conditions on Day 1 in treatment period 1, 2 and 3.
- Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet): Participants received a single oral dose of GSK3640254 / DTG, 150 mg/50 mg (1 bilayer tablet) FDC under moderate fat and calorie conditions on Day 1 in treatment period 1, 2 and 3.
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 18 | 20 | 16
Hours*microgram per milliliter | 22.13 (46.8) | 21.93 (36.6) | 22.63 (38.0)
Statistical Analysis 1: Comparison: Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg vs Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet); Test type: Other; Ratio of geometric Least Square mean = 1.025, 90% CI 2-sided [0.9335 to 1.126] — An analysis of variance with treatment, period, and sequence as fixed effects and participant nested within a sequence as a random effect was performed on the natural ln-transformed parameter AUC(0-inf)
Statistical Analysis 2: Comparison: Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg vs Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet); Test type: Other; Ratio of geometric Least Square mean = 1.072, 90% CI 2-sided [0.9693 to 1.185] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Part 1: Area Under the Plasma Concentration-time Curve From Time 0 to Time t (AUC[0-t]) of GSK3640254
Description: Blood samples were collected at indicated time points for PK analysis of GSK3640254.
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Hours*microgram per milliliter | 17.62 (55.4) | 19.14 (42.9) | 18.69 (42.4)
Statistical Analysis 1: Comparison: Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg vs Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet); Test type: Other; Ratio of geometric Least Square mean = 1.126, 90% CI 2-sided [0.9918 to 1.278] — An analysis of variance with treatment, period, and sequence as fixed effects and participant nested within a sequence as a random effect was performed on the natural ln-transformed parameter AUC(0-t)
Statistical Analysis 2: Comparison: Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg vs Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet); Test type: Other; Ratio of geometric Least Square mean = 1.055, 90% CI 2-sided [0.9278 to 1.201] — [estimate comment as in outcome 2, analysis 1]

3. Primary Outcome: Part 1: Maximum Observed Concentration (Cmax) of GSK3640254
Description: Blood samples were collected at indicated time points for PK analysis of GSK3640254.
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Microgram per milliliter | 0.7382 (40.3) | 0.7610 (33.5) | 0.7579 (40.1)
Statistical Analysis 1: Comparison: Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg vs Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet); Test type: Other; Ratio of geometric Least Square mean = 1.036, 90% CI 2-sided [0.9209 to 1.166] — An analysis of variance with treatment, period, and sequence as fixed effects and participant nested within a sequence as a random effect was performed on the natural ln-transformed parameter Cmax
Statistical Analysis 2: Comparison: Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg vs Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet); Test type: Other; Ratio of geometric Least Square mean = 1.020, 90% CI 2-sided [0.9049 to 1.151] — [estimate comment as in outcome 3, analysis 1]

4. Primary Outcome: Part 1: AUC(0-inf) of DTG
Description: Blood samples were collected at indicated time points for PK analysis of DTG.
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Hours*microgram per milliliter | 74.18 (30.7) | 82.13 (26.1) | 80.53 (34.7)
Statistical Analysis 1: Comparison: Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg vs Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet); Test type: Other; Ratio of geometric Least Square mean = 1.129, 90% CI 2-sided [1.067 to 1.195] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg vs Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet); Test type: Other; Ratio of geometric Least Square mean = 1.112, 90% CI 2-sided [1.050 to 1.178] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Part 1: AUC(0-t) of DTG
Description: Blood samples were collected at indicated time points for PK analysis of DTG.
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Hours*microgram per milliliter | 68.91 (32.5) | 77.89 (29.0) | 73.44 (37.0)
Statistical Analysis 1: Comparison: Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg vs Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet); Test type: Other; Ratio of geometric Least Square mean = 1.164, 90% CI 2-sided [1.070 to 1.267] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg vs Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet); Test type: Other; Ratio of geometric Least Square mean = 1.087, 90% CI 2-sided [0.9975 to 1.184] — [estimate comment as in outcome 2, analysis 1]

6. Primary Outcome: Part 1: Cmax of DTG
Description: Blood samples were collected at indicated time points for PK analysis of DTG.
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Microgram per milliliter | 4.182 (18.5) | 4.432 (17.8) | 4.264 (23.2)
Statistical Analysis 1: Comparison: Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg vs Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet); Test type: Other; Ratio of geometric Least Square mean = 1.078, 90% CI 2-sided [1.036 to 1.122] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg vs Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet); Test type: Other; Ratio of geometric Least Square mean = 1.032, 90% CI 2-sided [0.9914 to 1.075] — [estimate comment as in outcome 3, analysis 1]

7. Primary Outcome: Part 2: AUC(0-inf) of GSK3640254
Description: Blood samples were collected at indicated time points for PK analysis of GSK3640254.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Groups:
- Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed): Participants received Treatment D a single oral dose of selected bilayer FDC from Part 1 of GSK3640254/DTG, 150 mg/50 mg under high fat and calorie conditions on Day 1 in each treatment period.
- Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted): Participants received Treatment E a single oral dose of selected bilayer FDC from Part 1 GSK3640254/DTG, 150 mg/50 mg administered under fasted conditions on Day 1 in each treatment period.
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 13
Hours*microgram per milliliter | 21.39 (38.0) | 6.622 (77.4)
Statistical Analysis 1: Comparison: Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) vs Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted); Test type: Other; Ratio of geometric Least Square mean = 2.705, 90% CI 2-sided [2.135 to 3.427] — [estimate comment as in outcome 1, analysis 1]

8. Primary Outcome: Part 2: AUC(0-t) of GSK3640254
Description: Blood samples were collected at indicated time points for PK analysis of GSK3640254.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 13
Hours*microgram per milliliter | 19.33 (36.6) | 6.027 (78.8)
Statistical Analysis 1: Comparison: Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) vs Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted); Test type: Other; Ratio of geometric Least Square mean = 2.761, 90% CI 2-sided [2.160 to 3.527] — [estimate comment as in outcome 2, analysis 1]

9. Primary Outcome: Part 2: Cmax of GSK3640254
Description: Blood samples were collected at indicated time points for PK analysis of GSK3640254.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 13
Microgram per milliliter | 0.6093 (41.3) | 0.2193 (92.1)
Statistical Analysis 1: Comparison: Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) vs Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted); Test type: Other; Ratio of geometric Least Square mean = 2.498, 90% CI 2-sided [1.821 to 3.425] — [estimate comment as in outcome 3, analysis 1]

10. Primary Outcome: Part 2: AUC(0-inf) of DTG
Description: Blood samples were collected at indicated time points for PK analysis of DTG.
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Hours*microgram per milliliter | 85.07 (29.0) | 64.61 (31.5)
Statistical Analysis 1: Comparison: Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) vs Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted); Test type: Other; Ratio of geometric Least Square mean = 1.316, 90% CI 2-sided [1.193 to 1.451] — [estimate comment as in outcome 1, analysis 1]

11. Primary Outcome: Part 2: AUC(0-t) of DTG
Description: Blood samples were collected at indicated time points for PK analysis of DTG.
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Hours*microgram per milliliter | 83.18 (28.2) | 63.17 (31.0)
Statistical Analysis 1: Comparison: Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) vs Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted); Test type: Other; Ratio of geometric Least Square mean = 1.316, 90% CI 2-sided [1.193 to 1.452] — [estimate comment as in outcome 2, analysis 1]

12. Primary Outcome: Part 2: Cmax of DTG
Description: Blood samples were collected at indicated time points for PK analysis of DTG.
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Microgram per milliliter | 4.000 (21.1) | 3.273 (28.4)
Statistical Analysis 1: Comparison: Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) vs Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted); Test type: Other; Ratio of geometric Least Square mean = 1.232, 90% CI 2-sided [1.138 to 1.333] — [estimate comment as in outcome 3, analysis 1]

13. Secondary Outcome: Part 1: Number of Participants With Non-Serious Adverse Events (Non-SAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any serious adverse event that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or other situations as per medical or scientific judgment. Adverse events which were not Serious Adverse Events were considered as Non-Serious adverse events.
Time Frame: Up to 17 days
Population: Safety Population consisted of all participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Participants
  Non-SAEs | 0 | 0 | 1
  SAEs | 0 | 0 | 0

14. Secondary Outcome: Part 2: Number of Participants With Non-SAEs and SAEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any serious adverse event that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or other situations as per medical or scientific judgment. Adverse events which were not Serious Adverse Events were considered as Non-Serious adverse events.
Time Frame: Up to 9 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Participants
  Non-SAEs | 1 | 2
  SAEs | 0 | 0

15. Secondary Outcome: Part 1: Absolute Values for Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets
Description: Blood samples were collected to analyze the hematology parameters: basophils, eosinophils, lymphocytes, monocytes, neutrophils, and platelets. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
10^9 cells per liter
  Basophils, Baseline (Day -1) | 0.035 (0.0144) | 0.036 (0.0140) | 0.036 (0.0132)
  Basophils, Day 2: number analyzed (Participants) | 21 | 21 | 20
  Basophils, Day 2 | 0.036 (0.0133) | 0.036 (0.0120) | 0.037 (0.0184)
  Basophils, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Basophils, Day 5 | 0.045 (0.0138) | 0.035 (0.0187) | 0.028 (0.0117)
  Basophils, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Basophils, Day 7 | 0.033 (0.0142) | 0.040 (0.0108) | 0.038 (0.0169)
  Eosinophils, Baseline (Day -1) | 0.157 (0.1455) | 0.150 (0.1300) | 0.171 (0.1559)
  Eosinophils, Day 2: number analyzed (Participants) | 21 | 21 | 20
  Eosinophils, Day 2 | 0.157 (0.1382) | 0.146 (0.1229) | 0.170 (0.1482)
  Eosinophils, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Eosinophils, Day 5 | 0.197 (0.1481) | 0.182 (0.1512) | 0.120 (0.1210)
  Eosinophils, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Eosinophils, Day 7 | 0.141 (0.1272) | 0.152 (0.1194) | 0.189 (0.1613)
  Lymphocytes, Baseline (Day -1) | 1.683 (0.3691) | 1.674 (0.2885) | 1.646 (0.3375)
  Lymphocytes, Day 2: number analyzed (Participants) | 21 | 21 | 20
  Lymphocytes, Day 2 | 1.647 (0.3715) | 1.735 (0.3019) | 1.711 (0.3950)
  Lymphocytes, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Lymphocytes, Day 5 | 1.835 (0.4113) | 1.663 (0.4034) | 1.705 (0.4574)
  Lymphocytes, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Lymphocytes, Day 7 | 1.630 (0.3049) | 1.675 (0.3398) | 1.592 (0.3674)
  Monocytes, Baseline (Day -1) | 0.396 (0.0834) | 0.396 (0.0878) | 0.419 (0.1464)
  Monocytes, Day 2: number analyzed (Participants) | 21 | 21 | 20
  Monocytes, Day 2 | 0.395 (0.0803) | 0.389 (0.0861) | 0.410 (0.0932)
  Monocytes, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Monocytes, Day 5 | 0.422 (0.0987) | 0.387 (0.0497) | 0.380 (0.1243)
  Monocytes, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Monocytes, Day 7 | 0.380 (0.0587) | 0.398 (0.1162) | 0.410 (0.0903)
  Neutrophils, Baseline (Day -1) | 2.729 (0.8510) | 2.691 (1.0455) | 2.906 (1.3028)
  Neutrophils, Day 2: number analyzed (Participants) | 21 | 21 | 20
  Neutrophils, Day 2 | 2.756 (0.8228) | 2.589 (0.9598) | 2.573 (0.9203)
  Neutrophils, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Neutrophils, Day 5 | 2.967 (0.8932) | 2.648 (0.8738) | 2.703 (2.0389)
  Neutrophils, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Neutrophils, Day 7 | 2.462 (0.9607) | 2.594 (1.1921) | 2.812 (0.9202)
  Platelets, Baseline (Day -1) | 247.8 (45.94) | 252.5 (52.73) | 256.5 (50.02)
  Platelets, Day 2: number analyzed (Participants) | 21 | 21 | 20
  Platelets, Day 2 | 254.6 (46.26) | 257.0 (54.66) | 260.4 (52.24)
  Platelets, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Platelets, Day 5 | 277.8 (35.13) | 268.7 (52.38) | 212.2 (44.62)
  Platelets, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Platelets, Day 7 | 237.9 (40.40) | 257.1 (55.49) | 271.4 (44.96)

16. Secondary Outcome: Part 2: Absolute Values for Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets
Description: Blood samples were collected to analyze the hematology parameters: basophils, eosinophils, lymphocytes, monocytes, neutrophils, leukocytes and platelets. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
10^9 cells per liter
  Basophils, Baseline (Day -1) | 0.046 (0.0289) | 0.041 (0.0242)
  Basophils, Day 2: number analyzed (Participants) | 16 | 18
  Basophils, Day 2 | 0.038 (0.0183) | 0.041 (0.0192)
  Basophils, Day 5: number analyzed (Participants) | 8 | 9
  Basophils, Day 5 | 0.051 (0.0253) | 0.037 (0.0141)
  Basophils, Day 7: number analyzed (Participants) | 9 | 9
  Basophils, Day 7 | 0.033 (0.0141) | 0.057 (0.0354)
  Eosinophils, Baseline (Day -1) | 0.128 (0.0688) | 0.138 (0.0880)
  Eosinophils, Day 2: number analyzed (Participants) | 16 | 18
  Eosinophils, Day 2 | 0.125 (0.0700) | 0.136 (0.0786)
  Eosinophils, Day 5: number analyzed (Participants) | 8 | 9
  Eosinophils, Day 5 | 0.131 (0.0869) | 0.111 (0.0601)
  Eosinophils, Day 7: number analyzed (Participants) | 9 | 9
  Eosinophils, Day 7 | 0.123 (0.0726) | 0.133 (0.0652)
  Lymphocytes, Baseline (Day -1) | 1.786 (0.4445) | 1.771 (0.4902)
  Lymphocytes, Day 2: number analyzed (Participants) | 16 | 18
  Lymphocytes, Day 2 | 1.884 (0.4805) | 1.838 (0.4761)
  Lymphocytes, Day 5: number analyzed (Participants) | 8 | 9
  Lymphocytes, Day 5 | 1.663 (0.5135) | 1.750 (0.3384)
  Lymphocytes, Day 7: number analyzed (Participants) | 9 | 9
  Lymphocytes, Day 7 | 1.827 (0.3937) | 1.730 (0.5080)
  Monocytes, Baseline (Day -1) | 0.466 (0.1086) | 0.443 (0.1100)
  Monocytes, Day 2: number analyzed (Participants) | 16 | 18
  Monocytes, Day 2 | 0.452 (0.1114) | 0.458 (0.1070)
  Monocytes, Day 5: number analyzed (Participants) | 8 | 9
  Monocytes, Day 5 | 0.479 (0.1512) | 0.430 (0.1021)
  Monocytes, Day 7: number analyzed (Participants) | 9 | 9
  Monocytes, Day 7 | 0.452 (0.0987) | 0.469 (0.1102)
  Neutrophils, Baseline (Day -1) | 3.094 (1.1911) | 3.138 (1.1817)
  Neutrophils, Day 2: number analyzed (Participants) | 16 | 18
  Neutrophils, Day 2 | 2.999 (1.1184) | 3.122 (1.1220)
  Neutrophils, Day 5: number analyzed (Participants) | 8 | 9
  Neutrophils, Day 5 | 3.891 (2.1672) | 3.234 (1.3698)
  Neutrophils, Day 7: number analyzed (Participants) | 9 | 9
  Neutrophils, Day 7 | 2.967 (1.0973) | 3.083 (1.1599)
  Platelets, Baseline (Day -1) | 291.6 (53.57) | 292.7 (59.84)
  Platelets, Day 2: number analyzed (Participants) | 16 | 18
  Platelets, Day 2 | 302.0 (56.30) | 299.7 (62.53)
  Platelets, Day 5: number analyzed (Participants) | 8 | 9
  Platelets, Day 5 | 278.6 (61.63) | 314.1 (53.97)
  Platelets, Day 7: number analyzed (Participants) | 9 | 9
  Platelets, Day 7 | 307.4 (55.38) | 274.4 (61.27)

17. Secondary Outcome: Part 1: Absolute Values for Hematology Parameter: Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Grams per liter
  Baseline (Day -1) | 139.8 (16.04) | 142.7 (16.64) | 138.8 (16.55)
  Day 2: number analyzed (Participants) | 21 | 21 | 20
  Day 2 | 141.1 (15.57) | 143.1 (15.14) | 139.2 (16.11)
  Day 5: number analyzed (Participants) | 6 | 6 | 6
  Day 5 | 134.8 (14.74) | 135.0 (15.19) | 141.8 (14.89)
  Day 7: number analyzed (Participants) | 11 | 13 | 10
  Day 7 | 145.8 (14.97) | 140.6 (18.11) | 138.1 (16.11)

18. Secondary Outcome: Part 2: Absolute Values for Hematology Parameter: Hemoglobin
Description: as for outcome 17
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Grams per liter
  Baseline (Day -1) | 139.8 (15.66) | 138.4 (14.09)
  Day 2: number analyzed (Participants) | 16 | 18
  Day 2 | 141.0 (15.86) | 140.7 (16.62)
  Day 5: number analyzed (Participants) | 8 | 9
  Day 5 | 143.1 (11.22) | 135.6 (18.04)
  Day 7: number analyzed (Participants) | 9 | 9
  Day 7 | 134.3 (15.82) | 144.2 (11.11)

19. Secondary Outcome: Part 1: Absolute Values for Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular volume. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Femtoliter
  Baseline (Day -1) | 86.45 (4.446) | 86.33 (4.376) | 86.94 (4.244)
  Day 2: number analyzed (Participants) | 21 | 21 | 20
  Day 2 | 86.26 (4.324) | 86.51 (4.392) | 86.99 (4.171)
  Day 5: number analyzed (Participants) | 6 | 6 | 6
  Day 5 | 86.48 (4.642) | 86.08 (4.923) | 87.58 (4.668)
  Day 7: number analyzed (Participants) | 11 | 13 | 10
  Day 7 | 86.12 (4.256) | 87.28 (4.120) | 86.09 (4.703)

20. Secondary Outcome: Part 2: Absolute Values for Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: as for outcome 19
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Femtoliter
  Baseline (Day -1) | 84.55 (5.141) | 84.89 (4.925)
  Day 2: number analyzed (Participants) | 16 | 18
  Day 2 | 84.30 (4.926) | 84.74 (5.146)
  Day 5: number analyzed (Participants) | 8 | 9
  Day 5 | 84.33 (3.593) | 84.50 (6.116)
  Day 7: number analyzed (Participants) | 9 | 9
  Day 7 | 84.37 (5.841) | 85.29 (4.042)

21. Secondary Outcome: Part 1: Absolute Values for Hematology Parameter: Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
10^12 cells per liter
  Baseline (Day -1) | 4.757 (0.4773) | 4.850 (0.5190) | 4.686 (0.4967)
  Day 2: number analyzed (Participants) | 21 | 21 | 20
  Day 2 | 4.822 (0.4863) | 4.855 (0.4740) | 4.700 (0.4353)
  Day 5: number analyzed (Participants) | 6 | 6 | 6
  Day 5 | 4.658 (0.4331) | 4.558 (0.3547) | 4.710 (0.5284)
  Day 7: number analyzed (Participants) | 11 | 13 | 10
  Day 7 | 4.939 (0.5032) | 4.752 (0.5521) | 4.700 (0.4412)

22. Secondary Outcome: Part 2: Absolute Values for Hematology Parameter: Erythrocytes
Description: as for outcome 21
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
10^12 cells per liter
  Baseline (Day -1) | 4.914 (0.5070) | 4.853 (0.5060)
  Day 2: number analyzed (Participants) | 16 | 18
  Day 2 | 4.958 (0.4930) | 4.913 (0.5727)
  Day 5: number analyzed (Participants) | 8 | 9
  Day 5 | 4.976 (0.4861) | 4.787 (0.4171)
  Day 7: number analyzed (Participants) | 9 | 9
  Day 7 | 4.760 (0.5021) | 4.942 (0.5117)

23. Secondary Outcome: Part 1: Absolute Values for Hematology Parameters: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Proportion of red blood cells in blood
  Baseline (Day -1) | 0.4110 (0.04343) | 0.4181 (0.04561) | 0.4070 (0.04490)
  Day 2: number analyzed (Participants) | 21 | 21 | 20
  Day 2 | 0.4156 (0.04297) | 0.4195 (0.04087) | 0.4087 (0.04260)
  Day 5: number analyzed (Participants) | 6 | 6 | 6
  Day 5 | 0.4025 (0.03930) | 0.3922 (0.03854) | 0.4117 (0.04206)
  Day 7: number analyzed (Participants) | 11 | 13 | 10
  Day 7 | 0.4246 (0.04202) | 0.4144 (0.04936) | 0.4047 (0.04553)

24. Secondary Outcome: Part 2: Absolute Values for Hematology Parameters: Hematocrit
Description: as for outcome 23
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Proportion of red blood cells in blood
  Baseline (Day -1) | 0.4145 (0.04184) | 0.4106 (0.03687)
  Day 2: number analyzed (Participants) | 16 | 18
  Day 2 | 0.4173 (0.04269) | 0.4153 (0.04510)
  Day 5: number analyzed (Participants) | 8 | 9
  Day 5 | 0.4183 (0.03167) | 0.4044 (0.04641)
  Day 7: number analyzed (Participants) | 9 | 9
  Day 7 | 0.4004 (0.04078) | 0.4201 (0.03113)

25. Secondary Outcome: Part 1: Absolute Values for Hematology Parameters: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Picograms
  Baseline (Day -1) | 29.37 (1.743) | 29.47 (1.859) | 29.65 (1.819)
  Day 2: number analyzed (Participants) | 21 | 21 | 20
  Day 2 | 29.28 (1.811) | 29.51 (1.834) | 29.63 (1.823)
  Day 5: number analyzed (Participants) | 6 | 6 | 6
  Day 5 | 28.95 (2.117) | 29.63 (2.113) | 30.23 (2.111)
  Day 7: number analyzed (Participants) | 11 | 13 | 10
  Day 7 | 29.61 (1.924) | 29.61 (1.853) | 29.34 (1.735)

26. Secondary Outcome: Part 2: Absolute Values for Hematology Parameters: Erythrocytes Mean Corpuscular Hemoglobin
Description: as for outcome 25
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Picograms
  Baseline (Day -1) | 28.51 (2.271) | 28.62 (2.379)
  Day 2: number analyzed (Participants) | 16 | 18
  Day 2 | 28.49 (2.208) | 28.68 (2.266)
  Day 5: number analyzed (Participants) | 8 | 9
  Day 5 | 28.84 (1.508) | 28.32 (2.810)
  Day 7: number analyzed (Participants) | 9 | 9
  Day 7 | 28.32 (2.878) | 29.27 (1.665)

27. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets
Description: Blood samples were collected to analyze the hematology parameters: basophils, eosinophils, lymphocytes, monocytes, neutrophils, and platelets. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 21 | 21 | 20
10^9 cells per liter
  Basophils, Day 2 | 0.000 (0.0112) | 0.000 (0.0128) | 0.002 (0.0114)
  Basophils, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Basophils, Day 5 | 0.003 (0.0137) | 0.002 (0.0117) | -0.007 (0.0121)
  Basophils, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Basophils, Day 7 | 0.002 (0.0075) | 0.002 (0.0109) | 0.006 (0.0117)
  Eosinophils, Day 2 | -0.005 (0.0340) | -0.004 (0.0393) | -0.001 (0.0253)
  Eosinophils, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Eosinophils, Day 5 | 0.012 (0.0722) | -0.020 (0.0379) | -0.022 (0.0739)
  Eosinophils, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Eosinophils, Day 7 | 0.006 (0.0437) | 0.013 (0.0632) | -0.015 (0.0450)
  Lymphocytes, Day 2 | -0.006 (0.2568) | 0.061 (0.1626) | 0.065 (0.1831)
  Lymphocytes, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Lymphocytes, Day 5 | 0.012 (0.2670) | -0.103 (0.2293) | 0.053 (0.5253)
  Lymphocytes, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Lymphocytes, Day 7 | -0.023 (0.1443) | 0.069 (0.2843) | 0.031 (0.2409)
  Monocytes, Day 2 | 0.000 (0.0662) | -0.008 (0.0650) | -0.009 (0.1268)
  Monocytes, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Monocytes, Day 5 | -0.022 (0.0679) | 0.000 (0.0672) | 0.012 (0.0286)
  Monocytes, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Monocytes, Day 7 | -0.006 (0.0585) | -0.005 (0.0901) | -0.044 (0.1607)
  Neutrophils, Day 2 | 0.000 (0.6401) | -0.103 (0.6015) | -0.334 (0.9923)
  Neutrophils, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Neutrophils, Day 5 | 0.092 (0.4511) | 0.007 (0.1939) | 0.222 (1.1719)
  Neutrophils, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Neutrophils, Day 7 | -0.269 (0.6770) | -0.066 (0.6836) | -0.642 (1.3252)
  Platelets, Day 2 | 4.4 (9.28) | 4.5 (15.78) | 4.0 (14.96)
  Platelets, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Platelets, Day 5 | 5.2 (13.27) | -1.5 (15.06) | -7.5 (16.21)
  Platelets, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Platelets, Day 7 | -2.2 (20.03) | 7.9 (26.01) | 3.1 (32.56)

28. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets
Description: as for outcome 27
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 16 | 18
10^9 cells per liter
  Basophils, Day 2 | -0.004 (0.0121) | -0.001 (0.0111)
  Basophils, Day 5: number analyzed (Participants) | 8 | 9
  Basophils, Day 5 | -0.010 (0.0200) | 0.003 (0.0071)
  Basophils, Day 7: number analyzed (Participants) | 9 | 9
  Basophils, Day 7 | 0.000 (0.0100) | 0.008 (0.0273)
  Eosinophils, Day 2 | -0.006 (0.0234) | -0.002 (0.0342)
  Eosinophils, Day 5: number analyzed (Participants) | 8 | 9
  Eosinophils, Day 5 | -0.001 (0.0236) | -0.012 (0.0205)
  Eosinophils, Day 7: number analyzed (Participants) | 9 | 9
  Eosinophils, Day 7 | 0.000 (0.0260) | -0.020 (0.0400)
  Lymphocytes, Day 2 | 0.068 (0.2198) | 0.067 (0.1895)
  Lymphocytes, Day 5: number analyzed (Participants) | 8 | 9
  Lymphocytes, Day 5 | -0.075 (0.1507) | -0.077 (0.1678)
  Lymphocytes, Day 7: number analyzed (Participants) | 9 | 9
  Lymphocytes, Day 7 | -0.003 (0.2733) | 0.016 (0.1068)
  Monocytes, Day 2 | -0.023 (0.0422) | 0.014 (0.0497)
  Monocytes, Day 5: number analyzed (Participants) | 8 | 9
  Monocytes, Day 5 | -0.009 (0.1040) | -0.022 (0.0851)
  Monocytes, Day 7: number analyzed (Participants) | 9 | 9
  Monocytes, Day 7 | 0.006 (0.0923) | 0.034 (0.0706)
  Neutrophils, Day 2 | -0.077 (0.4373) | -0.016 (0.4117)
  Neutrophils, Day 5: number analyzed (Participants) | 8 | 9
  Neutrophils, Day 5 | 0.719 (1.2615) | 0.268 (0.8053)
  Neutrophils, Day 7: number analyzed (Participants) | 9 | 9
  Neutrophils, Day 7 | -0.058 (0.6203) | -0.226 (0.4835)
  Platelets, Day 2 | 6.1 (16.69) | 7.1 (12.62)
  Platelets, Day 5: number analyzed (Participants) | 8 | 9
  Platelets, Day 5 | 0.0 (7.19) | 6.7 (11.32)
  Platelets, Day 7: number analyzed (Participants) | 9 | 9
  Platelets, Day 7 | 4.2 (29.94) | -3.4 (30.53)

29. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 21 | 21 | 20
Grams per liter
  Day 2 | 1.2 (5.98) | 0.4 (5.44) | 0.4 (5.09)
  Day 5: number analyzed (Participants) | 6 | 6 | 6
  Day 5 | 0.5 (4.46) | -2.7 (4.59) | -1.3 (5.01)
  Day 7: number analyzed (Participants) | 11 | 13 | 10
  Day 7 | -1.8 (3.16) | -3.2 (7.57) | 0.0 (5.10)

30. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Hemoglobin
Description: as for outcome 29
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 16 | 18
Grams per liter
  Day 2 | 1.4 (4.86) | 2.2 (4.66)
  Day 5: number analyzed (Participants) | 8 | 9
  Day 5 | -1.4 (4.00) | 1.2 (5.52)
  Day 7: number analyzed (Participants) | 9 | 9
  Day 7 | -1.2 (4.35) | 1.7 (3.84)

31. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular volume. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 21 | 21 | 20
Femtoliter
  Day 2 | -0.06 (0.576) | 0.18 (0.658) | 0.05 (0.664)
  Day 5: number analyzed (Participants) | 6 | 6 | 6
  Day 5 | 0.32 (0.615) | 0.42 (0.611) | 0.13 (0.423)
  Day 7: number analyzed (Participants) | 11 | 13 | 10
  Day 7 | -0.58 (0.456) | 0.10 (0.663) | -0.09 (0.780)

32. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: as for outcome 31
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 16 | 18
Femtoliter
  Day 2 | -0.05 (0.629) | -0.16 (0.444)
  Day 5: number analyzed (Participants) | 8 | 9
  Day 5 | -0.31 (0.479) | 0.13 (0.552)
  Day 7: number analyzed (Participants) | 9 | 9
  Day 7 | -0.11 (0.992) | -0.13 (0.418)

33. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameter: Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 21 | 21 | 20
10^12 cells per liter
  Day 2 | 0.052 (0.1937) | 0.005 (0.1651) | 0.014 (0.1672)
  Day 5: number analyzed (Participants) | 6 | 6 | 6
  Day 5 | 0.020 (0.1642) | -0.097 (0.1592) | -0.062 (0.1297)
  Day 7: number analyzed (Participants) | 11 | 13 | 10
  Day 7 | -0.043 (0.1286) | -0.115 (0.2308) | 0.010 (0.2011)

34. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Erythrocytes
Description: as for outcome 33
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 16 | 18
10^12 cells per liter
  Day 2 | 0.034 (0.1628) | 0.061 (0.1886)
  Day 5: number analyzed (Participants) | 8 | 9
  Day 5 | -0.024 (0.1464) | 0.027 (0.2285)
  Day 7: number analyzed (Participants) | 9 | 9
  Day 7 | -0.077 (0.1875) | -0.003 (0.1151)

35. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hemotocrit. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 21 | 21 | 20
Proportion of red blood cells in blood
  Day 2 | 0.0042 (0.01656) | 0.0013 (0.01405) | 0.0017 (0.01477)
  Day 5: number analyzed (Participants) | 6 | 6 | 6
  Day 5 | 0.0027 (0.01253) | -0.0067 (0.01369) | -0.0048 (0.01148)
  Day 7: number analyzed (Participants) | 11 | 13 | 10
  Day 7 | -0.0066 (0.01184) | -0.0092 (0.01971) | 0.0011 (0.01930)

36. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameters: hemotocrit. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 16 | 18
Proportion of red blood cells in blood
  Day 2 | 0.0029 (0.01474) | 0.0047 (0.01576)
  Day 5: number analyzed (Participants) | 8 | 9
  Day 5 | -0.0038 (0.01403) | 0.0040 (0.02060)
  Day 7: number analyzed (Participants) | 9 | 9
  Day 7 | -0.0074 (0.01795) | -0.0007 (0.01093)

37. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Days 2, 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 21 | 21 | 20
Picograms
  Day 2 | -0.02 (0.319) | 0.04 (0.368) | -0.02 (0.233)
  Day 5: number analyzed (Participants) | 6 | 6 | 6
  Day 5 | 0.05 (0.138) | 0.07 (0.280) | 0.17 (0.301)
  Day 7: number analyzed (Participants) | 11 | 13 | 10
  Day 7 | -0.05 (0.372) | 0.01 (0.423) | -0.16 (0.320)

38. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: as for outcome 37
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 16 | 18
Picograms
  Day 2 | 0.07 (0.451) | 0.06 (0.463)
  Day 5: number analyzed (Participants) | 8 | 9
  Day 5 | -0.13 (0.255) | 0.00 (0.387)
  Day 7: number analyzed (Participants) | 9 | 9
  Day 7 | 0.21 (0.483) | 0.34 (0.445)

39. Secondary Outcome: Part 1: Absolute Values for Clinical Chemistry Parameters: Alanine Amino Transferase (ALT), Alkaline Phosphatase (ALP), Aspartate Amino Transferase (AST), Gamma Glutamyl Transferase (GGT), Lactate Dehydrogenase (LDH), Creatinine Kinase (CK)
Description: Blood samples were collected to analyze the chemistry parameters: ALT, ALP, AST, GGT, LDH, CK. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1), and Days 2, 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
International units per Liter
  ALT, Baseline (Day -1) | 16.4 (9.44) | 19.1 (13.65) | 18.9 (15.33)
  ALT, Day 2 | 16.3 (9.32) | 17.4 (9.99) | 18.4 (12.29)
  ALT, Day 5: number analyzed (Participants) | 6 | 6 | 6
  ALT, Day 5 | 14.0 (4.56) | 16.7 (8.64) | 19.5 (16.67)
  ALT, Day 7: number analyzed (Participants) | 11 | 13 | 10
  ALT, Day 7 | 20.5 (14.81) | 20.8 (18.34) | 17.2 (9.60)
  ALP, Baseline (Day -1) | 54.6 (14.90) | 55.6 (15.14) | 53.4 (15.34)
  ALP, Day 2 | 56.5 (14.72) | 57.6 (14.03) | 55.2 (15.58)
  ALP, Day 5: number analyzed (Participants) | 6 | 6 | 6
  ALP, Day 5 | 49.8 (13.69) | 60.8 (12.62) | 53.8 (17.62)
  ALP, Day 7: number analyzed (Participants) | 11 | 13 | 10
  ALP, Day 7 | 55.1 (14.74) | 52.8 (16.34) | 59.3 (16.35)
  AST, Baseline (Day -1) | 16.3 (4.84) | 17.0 (5.63) | 17.1 (6.23)
  AST, Day 2 | 15.8 (4.02) | 16.1 (4.57) | 17.1 (5.92)
  AST, Day 5: number analyzed (Participants) | 6 | 6 | 6
  AST, Day 5 | 14.8 (4.26) | 16.2 (4.92) | 16.3 (2.07)
  AST, Day 7: number analyzed (Participants) | 11 | 13 | 10
  AST, Day 7 | 16.5 (5.13) | 17.5 (7.31) | 17.5 (6.19)
  GGT, Baseline (Day -1) | 22.1 (15.68) | 22.9 (16.21) | 22.2 (15.53)
  GGT, Day 2 | 22.0 (14.57) | 22.8 (15.45) | 22.7 (13.77)
  GGT, Day 5: number analyzed (Participants) | 6 | 6 | 6
  GGT, Day 5 | 22.3 (19.38) | 21.8 (6.11) | 20.5 (12.36)
  GGT, Day 7: number analyzed (Participants) | 11 | 13 | 10
  GGT, Day 7 | 21.4 (10.08) | 22.9 (18.60) | 26.8 (20.97)
  LDH, Baseline (Day -1) | 121.7 (19.59) | 121.0 (24.41) | 119.5 (22.30)
  LDH, Day 2 | 119.1 (16.92) | 120.1 (23.02) | 123.5 (25.15)
  LDH, Day 5: number analyzed (Participants) | 6 | 6 | 6
  LDH, Day 5 | 119.5 (15.54) | 114.0 (21.22) | 107.5 (16.08)
  LDH, Day 7: number analyzed (Participants) | 11 | 13 | 10
  LDH, Day 7 | 105.3 (12.41) | 118.1 (22.72) | 116.0 (20.23)
  CK, Baseline (Day -1) | 101.0 (49.01) | 115.1 (114.93) | 106.8 (93.82)
  CK, Day 2 | 89.7 (51.73) | 104.8 (109.70) | 107.0 (114.66)
  CK, Day 5: number analyzed (Participants) | 6 | 6 | 6
  CK, Day 5 | 69.0 (33.00) | 96.5 (63.32) | 85.8 (40.74)
  CK, Day 7: number analyzed (Participants) | 11 | 13 | 10
  CK, Day 7 | 90.8 (51.77) | 104.6 (109.85) | 88.2 (46.19)

40. Secondary Outcome: Part 2: Absolute Values of Clinical Chemistry Parameters: ALT, ALP, AST, GGT, LDH, CK
Description: as for outcome 39
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
International units per Liter
  ALT, Baseline (Day -1) | 18.9 (12.42) | 18.8 (13.37)
  ALT, Day 2: number analyzed (Participants) | 16 | 18
  ALT, Day 2 | 18.6 (11.57) | 18.9 (12.65)
  ALT, Day 5: number analyzed (Participants) | 8 | 9
  ALT, Day 5 | 18.5 (11.82) | 25.2 (20.47)
  ALT, Day 7: number analyzed (Participants) | 9 | 9
  ALT, Day 7 | 21.8 (16.34) | 18.1 (9.97)
  ALP Baseline (Day -1) | 63.2 (18.86) | 61.6 (18.57)
  ALP, Day 2: number analyzed (Participants) | 16 | 18
  ALP, Day 2 | 62.1 (18.43) | 62.1 (18.75)
  ALP, Day 5: number analyzed (Participants) | 8 | 9
  ALP, Day 5 | 61.6 (18.18) | 70.4 (21.18)
  ALP, Day 7: number analyzed (Participants) | 9 | 9
  ALP, Day 7 | 66.6 (17.59) | 58.8 (19.73)
  AST, Baseline (Day -1) | 16.4 (4.15) | 16.7 (4.92)
  AST, Day 2: number analyzed (Participants) | 16 | 18
  AST, Day 2 | 15.6 (3.36) | 16.1 (4.30)
  AST, Day 5: number analyzed (Participants) | 8 | 9
  AST, Day 5 | 17.0 (2.88) | 20.1 (7.79)
  AST, Day 7: number analyzed (Participants) | 9 | 9
  AST, Day 7 | 17.7 (6.56) | 15.9 (2.71)
  GGT, Baseline (Day -1) | 21.6 (8.81) | 21.7 (9.34)
  GGT, Day 2: number analyzed (Participants) | 16 | 18
  GGT, Day 2 | 20.9 (8.62) | 22.2 (9.67)
  GGT, Day 5: number analyzed (Participants) | 8 | 9
  GGT, Day 5 | 21.6 (8.33) | 22.8 (11.91)
  GGT, Day 7: number analyzed (Participants) | 9 | 9
  GGT, Day 7 | 20.8 (9.65) | 21.8 (8.30)
  LDH, Baseline (Day -1) | 125.5 (14.23) | 123.4 (14.62)
  LDH, Day 2: number analyzed (Participants) | 16 | 18
  LDH, Day 2 | 117.8 (13.32) | 118.4 (11.64)
  LDH, Day 5: number analyzed (Participants) | 8 | 9
  LDH, Day 5 | 122.6 (16.59) | 122.6 (14.56)
  LDH, Day 7: number analyzed (Participants) | 9 | 9
  LDH, Day 7 | 119.2 (14.92) | 124.9 (17.95)
  CK, Baseline (Day -1) | 101.8 (52.32) | 103.3 (56.84)
  CK, Day 2: number analyzed (Participants) | 16 | 18
  CK, Day 2 | 89.5 (45.43) | 89.9 (41.11)
  CK, Day 5: number analyzed (Participants) | 8 | 9
  CK, Day 5 | 95.8 (38.31) | 99.8 (65.97)
  CK, Day 7: number analyzed (Participants) | 9 | 9
  CK, Day 7 | 97.7 (65.84) | 85.9 (31.47)

41. Secondary Outcome: Part 1: Absolute Values of Clinical Chemistry Parameters: Calcium, Carbon-dioxide (CO2), Chloride, Glucose, Potassium, Sodium, Urea Nitrogen, Phosphorus, Triglycerides, Cholesterol, and Anion Gap
Description: Blood samples were collected to analyze the chemistry parameters: calcium, CO2, chloride, glucose, potassium, sodium, urea nitrogen, phosphorus, triglycerides, cholesterol, and anion gap. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1), and Days 2, 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Millimoles per liter
  Calcium, Baseline (Day -1) | 2.357 (0.0999) | 2.366 (0.1034) | 2.347 (0.0839)
  Calcium, Day 2 | 2.371 (0.0986) | 2.377 (0.0868) | 2.379 (0.1009)
  Calcium, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Calcium, Day 5 | 2.345 (0.0948) | 2.407 (0.0509) | 2.393 (0.1171)
  Calcium, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Calcium, Day 7 | 2.380 (0.0949) | 2.348 (0.1014) | 2.371 (0.1201)
  CO2, Baseline (Day -1) | 30.5 (1.90) | 30.2 (2.14) | 30.3 (1.83)
  CO2, Day 2 | 29.4 (2.24) | 29.8 (2.12) | 29.8 (2.36)
  CO2, Day 5: number analyzed (Participants) | 6 | 6 | 6
  CO2, Day 5 | 28.2 (1.94) | 29.3 (2.34) | 29.7 (2.50)
  CO2, Day 7: number analyzed (Participants) | 11 | 13 | 10
  CO2, Day 7 | 30.5 (2.50) | 30.5 (1.98) | 30.0 (2.05)
  Chloride, Baseline (Day -1) | 101.7 (1.49) | 101.8 (2.07) | 102.1 (2.21)
  Chloride, Day 2 | 102.0 (2.53) | 101.6 (2.11) | 102.0 (2.32)
  Chloride, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Chloride, Day 5 | 102.8 (1.47) | 101.3 (2.16) | 101.7 (1.86)
  Chloride, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Chloride, Day 7 | 101.9 (1.92) | 102.4 (2.02) | 101.8 (1.03)
  Glucose, Baseline (Day -1) | 5.125 (0.4472) | 5.114 (0.3745) | 5.074 (0.3816)
  Glucose, Day 2 | 4.927 (0.4659) | 4.979 (0.4960) | 4.813 (0.4044)
  Glucose, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Glucose, Day 5 | 4.643 (0.3725) | 5.153 (0.3527) | 5.123 (0.4912)
  Glucose, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Glucose, Day 7 | 5.207 (0.3982) | 4.980 (0.4112) | 4.946 (0.3303)
  Potassium, Baseline (Day -1) | 4.20 (0.233) | 4.30 (4.24) | 4.24 (0.315)
  Potassium, Day 2 | 4.22 (0.246) | 4.12 (0.266) | 4.27 (0.334)
  Potassium, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Potassium, Day 5 | 4.18 (0.147) | 4.08 (0.271) | 4.15 (0.513)
  Potassium, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Potassium, Day 7 | 4.35 (0.383) | 4.24 (0.331) | 4.16 (0.165)
  Sodium, Baseline (Day -1) | 137.5 (2.48) | 137.9 (2.15) | 137.6 (2.37)
  Sodium, Day 2 | 137.5 (2.22) | 137.8 (1.73) | 137.9 (1.76)
  Sodium, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Sodium, Day 5 | 137.8 (1.83) | 137.2 (2.14) | 137.8 (2.64)
  Sodium, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Sodium, Day 7 | 138.2 (1.99) | 138.2 (2.20) | 137.2 (2.39)
  Urea nitrogen, Baseline (Day -1) | 4.105 (0.9931) | 4.398 (0.9260) | 4.216 (0.5976)
  Urea nitrogen, Day 2 | 4.625 (0.8713) | 4.731 (0.8265) | 4.491 (0.8115)
  Urea nitrogen, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Urea nitrogen, Day 5 | 3.980 (0.4246) | 4.378 (0.6674) | 4.368 (0.6707)
  Urea nitrogen, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Urea nitrogen, Day 7 | 4.810 (1.0170) | 4.220 (0.5511) | 4.439 (1.0769)
  Phosphate, Baseline (Day -1) | 1.126 (0.1429) | 1.095 (0.1602) | 1.156 (0.1414)
  Phosphate, Day 2 | 1.195 (0.1672) | 1.173 (0.1474) | 1.238 (0.1306)
  Phosphate, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Phosphate, Day 5 | 1.267 (0.1007) | 1.142 (0.2344) | 1.178 (0.1574)
  Phosphate, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Phosphate, Day 7 | 1.114 (0.0886) | 1.198 (0.1058) | 1.172 (0.1494)
  Triglycerides, Baseline (Day -1) | 1.161 (0.3495) | 1.284 (0.6031) | 1.011 (0.3381)
  Triglycerides, Day 2 | 1.255 (0.5400) | 1.271 (0.6676) | 1.022 (0.3455)
  Triglycerides, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Triglycerides, Day 5 | 0.907 (0.2482) | 1.020 (0.4494) | 0.827 (0.2523)
  Triglycerides Day 7: number analyzed (Participants) | 11 | 13 | 10
  Triglycerides Day 7 | 1.316 (0.6488) | 0.972 (0.3031) | 1.048 (0.3121)
  Cholesterol, Baseline (Day -1) | 4.666 (0.6505) | 4.737 (0.7591) | 4.674 (0.6908)
  Cholesterol, Day 2 | 4.783 (0.6972) | 4.795 (0.7617) | 4.726 (0.7404)
  Cholesterol, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Cholesterol, Day 5 | 4.863 (0.6029) | 4.507 (1.2255) | 4.292 (0.4032)
  Cholesterol, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Cholesterol, Day 7 | 4.415 (0.5871) | 4.776 (0.6017) | 4.590 (0.7417)
  Anion gap, Baseline (Day -1) | 9.5 (1.30) | 10.1 (1.62) | 9.6 (1.43)
  Anion gap, Day 2 | 10.3 (1.94) | 10.5 (1.29) | 10.3 (2.23)
  Anion gap, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Anion gap, Day 5 | 10.8 (1.72) | 10.7 (1.63) | 10.8 (1.72)
  Anion gap, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Anion gap, Day 7 | 10.2 (1.25) | 9.7 (1.38) | 9.4 (1.65)

42. Secondary Outcome: Part 2: Absolute Values of Clinical Chemistry Parameters: Calcium, CO2, Chloride, Glucose, Potassium, Sodium, Urea Nitrogen, Phosphorus, Triglycerides, Cholesterol, and Anion Gap
Description: as for outcome 41
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Millimoles per liter
  Calcium, Baseline (Day -1) | 2.356 (0.0947) | 2.354 (0.0833)
  Calcium, Day 2: number analyzed (Participants) | 16 | 18
  Calcium, Day 2 | 2.343 (0.0922) | 2.362 (0.0854)
  Calcium, Day 5: number analyzed (Participants) | 8 | 9
  Calcium, Day 5 | 2.315 (0.0991) | 2.381 (0.0764)
  Calcium, Day 7: number analyzed (Participants) | 9 | 9
  Calcium, Day 7 | 2.362 (0.1049) | 2.340 (0.0616)
  CO2, Baseline (Day -1) | 31.2 (1.42) | 31.1 (1.51)
  CO2, Day 2: number analyzed (Participants) | 16 | 18
  CO2, Day 2 | 29.8 (2.10) | 30.1 (2.10)
  CO2, Day 5: number analyzed (Participants) | 8 | 9
  CO2, Day 5 | 30.1 (1.64) | 30.8 (1.86)
  CO2, Day 7: number analyzed (Participants) | 9 | 9
  CO2, Day 7 | 31.3 (1.87) | 31.1 (1.17)
  Chloride, Baseline (Day -1) | 101.8 (2.11) | 102.1 (1.45)
  Chloride, Day 2: number analyzed (Participants) | 16 | 18
  Chloride, Day 2 | 102.3 (1.34) | 101.7 (1.64)
  Chloride, Day 5: number analyzed (Participants) | 8 | 9
  Chloride, Day 5 | 102.0 (1.93) | 101.4 (1.01)
  Chloride, Day 7: number analyzed (Participants) | 9 | 9
  Chloride, Day 7 | 102.3 (1.87) | 102.1 (2.20)
  Glucose, Baseline (Day -1) | 4.872 (0.3107) | 4.913 (0.3252)
  Glucose, Day 2: number analyzed (Participants) | 16 | 18
  Glucose, Day 2 | 4.784 (0.3470) | 4.989 (0.3379)
  Glucose, Day 5: number analyzed (Participants) | 8 | 9
  Glucose, Day 5 | 4.606 (0.3351) | 4.729 (0.1985)
  Glucose, Day 7: number analyzed (Participants) | 9 | 9
  Glucose, Day 7 | 4.984 (0.3691) | 4.754 (0.3304)
  Potassium, Baseline (Day -1) | 4.29 (0.183) | 4.27 (0.225)
  Potassium, Day 2: number analyzed (Participants) | 16 | 18
  Potassium, Day 2 | 4.30 (0.193) | 4.36 (0.350)
  Potassium, Day 5: number analyzed (Participants) | 8 | 9
  Potassium, Day 5 | 4.33 (0.369) | 4.18 (0.222)
  Potassium, Day 7: number analyzed (Participants) | 9 | 9
  Potassium, Day 7 | 4.26 (0.133) | 4.46 (0.364)
  Sodium, Baseline (Day -1) | 138.2 (2.02) | 138.1 (1.55)
  Sodium, Day 2: number analyzed (Participants) | 16 | 18
  Sodium, Day 2 | 137.8 (1.83) | 137.8 (2.39)
  Sodium, Day 5: number analyzed (Participants) | 8 | 9
  Sodium, Day 5 | 137.4 (1.69) | 138.1 (1.90)
  Sodium, Day 7: number analyzed (Participants) | 9 | 9
  Sodium, Day 7 | 138.9 (1.17) | 138.4 (2.40)
  Urea nitrogen, Baseline (Day -1) | 4.193 (0.9707) | 4.289 (0.8517)
  Urea nitrogen, Day 2: number analyzed (Participants) | 16 | 18
  Urea nitrogen, Day 2 | 4.511 (0.8025) | 4.917 (1.2215)
  Urea nitrogen, Day 5: number analyzed (Participants) | 8 | 9
  Urea nitrogen, Day 5 | 4.488 (0.7840) | 4.197 (0.9577)
  Urea nitrogen, Day 7: number analyzed (Participants) | 9 | 9
  Urea nitrogen, Day 7 | 4.130 (0.9850) | 4.889 (1.2618)
  Phosphate, Baseline (Day -1) | 1.129 (0.1711) | 1.137 (0.1644)
  Phosphate, Day 2: number analyzed (Participants) | 16 | 18
  Phosphate, Day 2 | 1.163 (0.1414) | 1.181 (0.1402)
  Phosphate, Day 5: number analyzed (Participants) | 8 | 9
  Phosphate, Day 5 | 1.149 (0.1183) | 1.159 (0.1837)
  Phosphate, Day 7: number analyzed (Participants) | 9 | 9
  Phosphate, Day 7 | 1.147 (0.1777) | 1.146 (0.1261)
  Triglycerides, Baseline (Day -1) | 1.380 (0.5675) | 1.346 (0.6796)
  Triglycerides, Day 2: number analyzed (Participants) | 16 | 18
  Triglycerides, Day 2 | 1.255 (0.5644) | 1.226 (0.4816)
  Triglycerides, Day 5: number analyzed (Participants) | 8 | 9
  Triglycerides, Day 5 | 1.268 (0.6846) | 1.044 (0.4087)
  Triglycerides, Day 7: number analyzed (Participants) | 9 | 9
  Triglycerides, Day 7 | 1.200 (0.5402) | 1.461 (0.7119)
  Cholesterol, Baseline (Day -1) | 4.477 (0.8449) | 4.454 (0.7606)
  Cholesterol, Day 2: number analyzed (Participants) | 16 | 18
  Cholesterol, Day 2 | 4.603 (0.7998) | 4.531 (0.8227)
  Cholesterol, Day 5: number analyzed (Participants) | 8 | 9
  Cholesterol, Day 5 | 4.591 (0.8199) | 4.287 (0.9845)
  Cholesterol, Day 7: number analyzed (Participants) | 9 | 9
  Cholesterol, Day 7 | 4.173 (0.7740) | 4.617 (0.8221)
  Anion Gap, Baseline (Day -1) | 9.5 (0.87) | 9.2 (0.92)
  Anion Gap, Day 2: number analyzed (Participants) | 16 | 18
  Anion Gap, Day 2 | 9.9 (0.85) | 10.4 (0.98)
  Anion Gap, Day 5: number analyzed (Participants) | 8 | 9
  Anion Gap, Day 5 | 9.6 (0.92) | 9.0 (2.83)
  Anion Gap, Day 7: number analyzed (Participants) | 9 | 9
  Anion Gap, Day 7 | 9.3 (0.87) | 9.6 (0.88)

43. Secondary Outcome: Part 1: Absolute Values for Chemistry Parameters: Serum Lipase, Serum Amylase
Description: Blood samples were collected to analyze the chemistry parameters: serum lipase and serum amylase. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1), and Days 2, 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per Liter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Units per Liter
  Serum lipase, Baseline (Day -1) | 32.5 (12.77) | 34.6 (17.45) | 31.1 (13.95)
  Serum lipase, Day 2 | 32.1 (13.07) | 40.4 (27.76) | 34.2 (13.50)
  Serum lipase, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Serum lipase, Day 5 | 34.3 (15.08) | 40.2 (19.87) | 27.7 (5.61)
  Serum lipase, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Serum lipase, Day 7 | 33.1 (17.23) | 28.8 (11.77) | 35.0 (17.18)
  Serum amylase, Baseline (Day -1) | 54.9 (13.67) | 58.9 (16.72) | 58.4 (14.51)
  Serum amylase, Day 2 | 58.9 (15.47) | 62.8 (18.88) | 61.7 (16.92)
  Serum amylase, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Serum amylase, Day 5 | 63.3 (9.91) | 55.2 (15.47) | 62.2 (23.16)
  Serum amylase, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Serum amylase, Day 7 | 62.0 (19.18) | 62.2 (14.71) | 56.2 (13.57)

44. Secondary Outcome: Part 2: Absolute Values for Chemistry Parameters: Serum Lipase, Serum Amylase
Description: Blood samples were collected to analyze the chemistry parameters: serum lipase, serum amylase. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per Liter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Units per Liter
  Serum lipase, Baseline (Day -1) | 32.1 (11.73) | 30.2 (10.22)
  Serum lipase, Day 2: number analyzed (Participants) | 16 | 18
  Serum lipase, Day 2 | 30.5 (11.60) | 30.4 (11.12)
  Serum lipase, Day 5: number analyzed (Participants) | 8 | 9
  Serum lipase, Day 5 | 28.6 (19.28) | 40.3 (15.17)
  Serum lipase, Day 7: number analyzed (Participants) | 9 | 9
  Serum lipase, Day 7 | 35.0 (6.22) | 25.2 (12.59)
  Serum amylase, Baseline (Day -1) | 58.7 (17.33) | 56.7 (15.19)
  Serum amylase, Day 2: number analyzed (Participants) | 16 | 18
  Serum amylase, Day 2 | 58.3 (17.08) | 58.8 (15.21)
  Serum amylase, Day 5: number analyzed (Participants) | 8 | 9
  Serum amylase, Day 5 | 53.9 (16.40) | 62.7 (14.06)
  Serum amylase, Day 7: number analyzed (Participants) | 9 | 9
  Serum amylase, Day 7 | 63.3 (15.98) | 51.7 (14.27)

45. Secondary Outcome: Part 1: Absolute Values of Clinical Chemistry Parameters: Albumin, Globulin and Protein
Description: Blood samples were collected to analyze the chemistry parameters: albumin, globulin and protein. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1), and Days 2, 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Grams per liter
  Albumin, Baseline (Day -1) | 43.8 (2.91) | 43.8 (3.12) | 43.8 (2.38)
  Albumin, Day 2 | 44.6 (2.61) | 44.5 (2.29) | 44.5 (2.46)
  Albumin, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Albumin, Day 5 | 43.8 (2.23) | 43.8 (2.32) | 43.2 (4.12)
  Albumin, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Albumin, Day 7 | 43.6 (2.66) | 43.9 (2.22) | 45.3 (2.16)
  Globulin, Baseline (Day -1) | 26.4 (4.04) | 27.0 (3.25) | 26.0 (3.63)
  Globulin, Day 2 | 27.3 (3.85) | 27.4 (3.72) | 27.1 (4.51)
  Globulin, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Globulin, Day 5 | 26.0 (2.61) | 28.0 (3.52) | 26.2 (3.37)
  Globulin, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Globulin, Day 7 | 27.1 (3.78) | 25.8 (3.60) | 25.9 (4.31)
  Protein, Baseline (Day -1) | 70.1 (5.10) | 70.8 (4.12) | 69.7 (4.46)
  Protein, Day 2 | 71.9 (4.86) | 71.9 (4.03) | 71.6 (5.60)
  Protein, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Protein, Day 5 | 69.8 (1.94) | 71.8 (4.71) | 69.3 (5.28)
  Protein, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Protein, Day 7 | 70.7 (4.90) | 69.8 (4.17) | 71.2 (4.71)

46. Secondary Outcome: Part 2: Absolute Values of Clinical Chemistry Parameters: Albumin, Globulin and Protein
Description: as for outcome 45
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Grams per liter
  Albumin, Baseline (Day -1) | 42.9 (3.72) | 43.1 (3.40)
  Albumin, Day 2: number analyzed (Participants) | 16 | 18
  Albumin, Day 2 | 43.3 (2.91) | 43.2 (3.26)
  Albumin, Day 5: number analyzed (Participants) | 8 | 9
  Albumin, Day 5 | 44.4 (2.56) | 44.9 (4.04)
  Albumin, Day 7: number analyzed (Participants) | 9 | 9
  Albumin, Day 7 | 43.3 (4.33) | 43.2 (2.39)
  Globulin, Baseline (Day -1) | 28.0 (3.39) | 27.2 (3.64)
  Globulin, Day 2: number analyzed (Participants) | 16 | 18
  Globulin, Day 2 | 28.5 (3.27) | 28.1 (3.47)
  Globulin, Day 5: number analyzed (Participants) | 8 | 9
  Globulin, Day 5 | 27.1 (3.94) | 30.4 (3.78)
  Globulin, Day 7: number analyzed (Participants) | 9 | 9
  Globulin, Day 7 | 28.4 (3.64) | 25.9 (3.48)
  Protein, Baseline (Day -1) | 70.9 (4.83) | 70.3 (4.69)
  Protein, Day 2: number analyzed (Participants) | 16 | 18
  Protein, Day 2 | 71.8 (3.60) | 71.3 (4.60)
  Protein, Day 5: number analyzed (Participants) | 8 | 9
  Protein, Day 5 | 71.5 (3.96) | 75.3 (5.00)
  Protein, Day 7: number analyzed (Participants) | 9 | 9
  Protein, Day 7 | 71.8 (6.04) | 69.1 (4.23)

47. Secondary Outcome: Part 1: Absolute Values of Clinical Chemistry Parameters: Creatinine, Direct Bilirubin, Bilirubin, and Urate
Description: Blood samples were collected to analyze the chemistry parameters: creatinine, direct bilirubin, bilirubin, urate. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1), and Days 2, 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Micromoles per liter
  Creatinine, Baseline (Day -1) | 74.58 (13.770) | 77.79 (14.328) | 75.32 (15.250)
  Creatinine, Day 2 | 82.89 (15.880) | 84.90 (17.025) | 81.47 (15.445)
  Creatinine, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Creatinine, Day 5 | 76.77 (9.046) | 77.20 (17.447) | 79.57 (18.646)
  Creatinine, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Creatinine, Day 7 | 82.05 (14.136) | 78.55 (15.613) | 74.53 (13.793)
  Direct bilirubin, Baseline (Day -1) | 1.93 (0.540) | 2.03 (0.597) | 2.03 (0.634)
  Direct bilirubin, Day 2 | 1.80 (0.532) | 1.97 (0.678) | 2.03 (0.687)
  Direct bilirubin, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Direct bilirubin, Day 5 | 1.67 (0.437) | 2.08 (0.694) | 2.28 (0.778)
  Direct bilirubin, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Direct bilirubin, Day 7 | 2.00 (0.548) | 1.88 (0.577) | 2.04 (0.648)
  Bilirubin, Baseline (Day -1) | 10.38 (3.283) | 11.43 (3.510) | 10.93 (3.805)
  Bilirubin, Day 2 | 9.70 (2.714) | 11.04 (3.619) | 10.72 (3.862)
  Bilirubin, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Bilirubin, Day 5 | 8.38 (3.021) | 9.95 (3.605) | 11.05 (3.553)
  Bilirubin, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Bilirubin, Day 7 | 10.92 (2.975) | 10.34 (3.510) | 10.11 (3.473)
  Urate, Baseline (Day -1) | 287.0 (67.20) | 291.8 (58.22) | 276.0 (58.76)
  Urate, Day 2 | 280.1 (64.07) | 283.9 (62.39) | 271.9 (54.52)
  Urate, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Urate, Day 5 | 235.0 (40.83) | 290.5 (53.91) | 292.3 (53.16)
  Urate, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Urate, Day 7 | 305.1 (55.55) | 271.8 (58.66) | 280.0 (53.36)

48. Secondary Outcome: Part 2: Absolute Values of Clinical Chemistry Parameters: Creatinine, Direct Bilirubin, Bilirubin, and Urate
Description: Blood samples were collected to analyze the chemistry parameters: creatinine, direct bilirubin, bilirubin, and urate. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Micromoles per liter
  Creatinine, Baseline (Day -1) | 81.02 (17.857) | 83.19 (19.817)
  Creatinine, Day 2: number analyzed (Participants) | 16 | 18
  Creatinine, Day 2 | 88.29 (21.603) | 90.17 (22.148)
  Creatinine, Day 5: number analyzed (Participants) | 8 | 9
  Creatinine, Day 5 | 85.31 (13.191) | 83.79 (24.894)
  Creatinine, Day 7: number analyzed (Participants) | 9 | 9
  Creatinine, Day 7 | 82.51 (25.513) | 82.90 (12.663)
  Direct bilirubin, Baseline (Day -1) | 1.71 (0.506) | 1.73 (0.470)
  Direct bilirubin, Day 2: number analyzed (Participants) | 16 | 18
  Direct bilirubin, Day 2 | 1.69 (0.431) | 1.77 (0.621)
  Direct bilirubin, Day 5: number analyzed (Participants) | 8 | 9
  Direct bilirubin, Day 5 | 1.89 (0.295) | 1.99 (0.851)
  Direct bilirubin, Day 7: number analyzed (Participants) | 9 | 9
  Direct bilirubin, Day 7 | 1.62 (0.565) | 1.72 (0.286)
  Bilirubin, Baseline (Day -1) | 9.64 (3.401) | 9.27 (2.548)
  Bilirubin, Day 2: number analyzed (Participants) | 16 | 18
  Bilirubin, Day 2 | 8.98 (1.548) | 9.58 (3.048)
  Bilirubin, Day 5: number analyzed (Participants) | 8 | 9
  Bilirubin, Day 5 | 9.55 (1.125) | 10.50 (5.312)
  Bilirubin, Day 7: number analyzed (Participants) | 9 | 9
  Bilirubin, Day 7 | 8.57 (3.324) | 9.90 (0.758)
  Urate, Baseline (Day -1) | 324.4 (66.68) | 329.2 (73.48)
  Urate, Day 2: number analyzed (Participants) | 16 | 18
  Urate, Day 2 | 307.0 (64.72) | 331.8 (81.70)
  Urate, Day 5: number analyzed (Participants) | 8 | 9
  Urate, Day 5 | 330.1 (68.86) | 306.0 (73.64)
  Urate, Day 7: number analyzed (Participants) | 9 | 9
  Urate, Day 7 | 308.0 (74.35) | 332.3 (62.07)

49. Secondary Outcome: Part 1: Change From Baseline in Chemistry Parameters: ALT, ALP, AST, GGT, LDH, CK
Description: Blood samples were collected to analyze the chemistry parameters: ALT, ALP, AST, GGT, LDH, CK. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Days 2, 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
International units per Liter
  ALT, Day 2 | -0.1 (2.49) | -1.7 (4.74) | -0.5 (5.50)
  ALT, Day 5: number analyzed (Participants) | 6 | 6 | 6
  ALT, Day 5 | -1.7 (4.37) | -0.2 (2.23) | -3.0 (8.39)
  ALT, Day 7: number analyzed (Participants) | 11 | 13 | 10
  ALT, Day 7 | 1.1 (5.97) | -0.3 (9.32) | 0.5 (7.93)
  ALP, Day 2 | 1.8 (5.14) | 2.0 (3.76) | 1.8 (4.66)
  ALP, Day 5: number analyzed (Participants) | 6 | 6 | 6
  ALP, Day 5 | -1.8 (3.25) | -1.0 (5.66) | -2.7 (6.74)
  ALP, Day 7: number analyzed (Participants) | 11 | 13 | 10
  ALP, Day 7 | 1.4 (3.67) | 0.8 (3.75) | 3.9 (5.55)
  AST, Day 2 | -0.5 (1.65) | -0.9 (2.32) | 0.0 (3.08)
  AST, Day 5: number analyzed (Participants) | 6 | 6 | 6
  AST, Day 5 | -2.0 (2.90) | 0.3 (1.63) | 0.0 (3.58)
  AST, Day 7: number analyzed (Participants) | 11 | 13 | 10
  AST, Day 7 | -0.4 (2.06) | -0.9 (3.62) | 0.6 (2.76)
  GGT, Day 2 | -0.1 (2.24) | 0.0 (1.43) | 0.6 (3.76)
  GGT, Day 5: number analyzed (Participants) | 6 | 6 | 6
  GGT, Day 5 | -3.0 (4.20) | -1.3 (1.86) | -1.0 (2.28)
  GGT, Day 7: number analyzed (Participants) | 11 | 13 | 10
  GGT, Day 7 | -0.1 (3.11) | -1.2 (2.48) | 2.4 (8.13)
  LDH, Day 2 | -2.6 (11.67) | -0.9 (10.41) | 4.0 (9.89)
  LDH, Day 5: number analyzed (Participants) | 6 | 6 | 6
  LDH, Day 5 | -16.5 (14.90) | 0.3 (7.26) | 2.2 (14.15)
  LDH, Day 7: number analyzed (Participants) | 11 | 13 | 10
  LDH, Day 7 | -8.8 (10.09) | -10.2 (9.54) | -5.3 (15.43)
  CK, Day 2 | -11.4 (33.22) | -10.3 (20.22) | 0.2 (27.16)
  CK, Day 5: number analyzed (Participants) | 6 | 6 | 6
  CK, Day 5 | -18.5 (20.66) | -1.8 (11.58) | 8.8 (13.75)
  CK, Day 7: number analyzed (Participants) | 11 | 13 | 10
  CK, Day 7 | -26.2 (43.88) | -27.3 (43.24) | -9.3 (22.62)

50. Secondary Outcome: Part 2: Change From Baseline in Chemistry Parameters: ALT, ALP, AST, GGT, LDH, CK
Description: as for outcome 49
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 16 | 18
International units per Liter
  ALT, Day 2 | -0.7 (3.48) | 0.1 (3.30)
  ALT, Day 5: number analyzed (Participants) | 8 | 9
  ALT, Day 5 | 1.1 (2.64) | 3.4 (7.21)
  ALT, Day 7: number analyzed (Participants) | 9 | 9
  ALT, Day 7 | 1.6 (5.77) | 2.2 (3.67)
  ALP, Day 2 | -0.1 (4.22) | 0.4 (3.65)
  ALP, Day 5: number analyzed (Participants) | 8 | 9
  ALP, Day 5 | 1.1 (3.56) | 3.9 (9.20)
  ALP, Day 7: number analyzed (Participants) | 9 | 9
  ALP, Day 7 | 1.0 (3.81) | 2.1 (4.26)
  AST, Day 2 | -0.8 (2.32) | -0.7 (1.81)
  AST, Day 5: number analyzed (Participants) | 8 | 9
  AST, Day 5 | 1.4 (1.06) | 2.4 (3.32)
  AST, Day 7: number analyzed (Participants) | 9 | 9
  AST, Day 7 | 0.7 (2.55) | 0.1 (1.69)
  GGT, Day 2 | -0.3 (1.08) | 0.5 (1.38)
  GGT, Day 5: number analyzed (Participants) | 8 | 9
  GGT, Day 5 | 0.9 (0.83) | 2.0 (3.67)
  GGT, Day 7: number analyzed (Participants) | 9 | 9
  GGT, Day 7 | -1.6 (3.09) | -0.9 (2.71)
  LDH, Day 2 | -7.1 (11.65) | -4.9 (8.68)
  LDH, Day 5: number analyzed (Participants) | 8 | 9
  LDH, Day 5 | -4.6 (10.89) | 3.3 (16.90)
  LDH, Day 7: number analyzed (Participants) | 9 | 9
  LDH, Day 7 | -4.8 (12.02) | -2.7 (11.92)
  CK, Day 2 | -6.9 (12.25) | -13.4 (20.32)
  CK, Day 5: number analyzed (Participants) | 8 | 9
  CK, Day 5 | 7.6 (11.56) | 2.1 (13.70)
  CK, Day 7: number analyzed (Participants) | 9 | 9
  CK, Day 7 | -16.3 (34.30) | -23.1 (36.97)

51. Secondary Outcome: Part 1: Change From Baseline in Clinical Chemistry Parameters: Calcium, CO2, Chloride, Glucose, Potassium, Sodium, Urea Nitrogen, Phosphorus, Triglycerides, Cholesterol, and Anion Gap
Description: Blood samples were collected to analyze the chemistry parameters: calcium, CO2, chloride, glucose, potassium, sodium, urea nitrogen, phosphorus, triglycerides, cholesterol, and anion gap. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Days 2, 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Millimoles per liter
  Calcium, Day 2 | 0.014 (0.0547) | 0.011 (0.0599) | 0.033 (0.0838)
  Calcium, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Calcium, Day 5 | -0.007 (0.0333) | 0.013 (0.0432) | 0.007 (0.0535)
  Calcium, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Calcium, Day 7 | 0.011 (0.0650) | -0.002 (0.0867) | 0.018 (0.0875)
  CO2, Day 2 | -1.1 (1.41) | -0.5 (1.33) | -0.5 (1.57)
  CO2, Day 5: number analyzed (Participants) | 6 | 6 | 6
  CO2, Day 5 | -1.7 (1.37) | -0.8 (1.17) | -1.7 (1.63)
  CO2, Day 7: number analyzed (Participants) | 11 | 13 | 10
  CO2, Day 7 | -0.5 (1.69) | 0.4 (2.22) | 0.0 (1.05)
  Chloride, Day 2 | 0.3 (1.94) | -0.1 (1.15) | -0.1 (1.47)
  Chloride, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Chloride, Day 5 | 1.7 (2.25) | -0.3 (1.03) | -1.5 (2.51)
  Chloride, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Chloride, Day 7 | 0.2 (1.89) | 0.8 (2.17) | -0.1 (2.23)
  Glucose, Day 2 | -0.197 (0.2209) | -0.135 (0.2856) | -0.262 (0.1809)
  Glucose, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Glucose, Day 5 | -0.093 (0.2550) | -0.035 (0.1792) | -0.105 (0.1735)
  Glucose, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Glucose, Day 7 | -0.086 (0.3962) | -0.066 (0.3024) | -0.171 (0.1920)
  Potassium, Day 2 | 0.02 (0.234) | -0.18 (0.274) | 0.03 (0.281)
  Potassium, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Potassium, Day 5 | 0.10 (0.290) | -0.05 (0.226) | -0.20 (0.369)
  Potassium, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Potassium, Day 7 | 0.10 (0.310) | -0.06 (0.198) | -0.08 (0.361)
  Sodium, Day 2 | 0.0 (1.95) | 1.64 (0.3) | 0.3 (2.24)
  Sodium, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Sodium, Day 5 | 1.0 (1.79) | -0.2 (1.17) | -1.3 (2.66)
  Sodium, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Sodium, Day 7 | -0.2 (2.36) | 0.4 (2.14) | -0.3 (2.31)
  Urea nitrogen, Day 2 | 0.520 (0.7073) | 0.333 (0.4752) | 0.4553 (0.4553)
  Urea nitrogen, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Urea nitrogen, Day 5 | 0.857 (0.4584) | 0.143 (0.5844) | -0.017 (0.6301)
  Urea nitrogen, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Urea nitrogen, Day 7 | 0.618 (0.7434) | -0.035 (0.5511) | 0.309 (0.7935)
  Phosphate, Day 2 | 0.069 (0.1242) | 0.078 (0.0972) | 0.082 (0.0716)
  Phosphate, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Phosphate, Day 5 | 0.082 (0.1232) | 0.048 (0.0952) | -0.002 (0.0964)
  Phosphate, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Phosphate, Day 7 | 0.036 (0.1218) | 0.099 (0.1245) | 0.052 (0.0487)
  Triglycerides, Day 2 | 0.095 (0.3467) | -0.013 (0.2499) | 0.011 (0.2280)
  Triglycerides, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Triglycerides, Day 5 | -0.192 (0.1338) | -0.223 (0.3551) | -0.185 (0.1778)
  Triglycerides, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Triglycerides, Day 7 | 0.160 (0.4290) | -0.149 (0.2656) | -0.016 (0.1888)
  Cholesterol, Day 2 | 0.117 (0.3551) | 0.058 (0.3115) | 0.052 (0.2865)
  Cholesterol, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Cholesterol, Day 5 | -0.098 (0.5254) | -0.022 (0.4323) | -0.252 (0.3485)
  Cholesterol, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Cholesterol, Day 7 | -0.033 (0.4137) | -0.137 (0.4751) | 0.056 (0.3841)
  Anion gap, Day 2 | 0.8 (2.07) | 0.3 (1.59) | 0.8 (2.36)
  Anion gap, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Anion gap, Day 5 | 1.0 (1.41) | 1.2 (1.17) | 1.7 (1.37)
  Anion gap, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Anion gap, Day 7 | 0.4 (1.29) | -0.8 (1.88) | -0.4 (1.35)

52. Secondary Outcome: Part 2: Change From Baseline in Clinical Chemistry Parameters: Calcium, CO2, Chloride, Glucose, Potassium, Sodium, Urea Nitrogen, Phosphorus, Triglycerides, Cholesterol, and Anion Gap
Description: as for outcome 51
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Millimoles per liter
  Calcium, Day 2: number analyzed (Participants) | 16 | 18
  Calcium, Day 2 | -0.008 (0.0764) | 0.007 (0.0585)
  Calcium, Day 5: number analyzed (Participants) | 8 | 9
  Calcium, Day 5 | -0.033 (0.0812) | 0.019 (0.0971)
  Calcium, Day 7: number analyzed (Participants) | 9 | 9
  Calcium, Day 7 | -0.002 (0.0814) | -0.007 (0.0779)
  CO2, Day 2: number analyzed (Participants) | 16 | 18
  CO2, Day 2 | -1.3 (1.49) | -1.0 (1.37)
  CO2, Day 5: number analyzed (Participants) | 8 | 9
  CO2, Day 5 | -1.1 (0.99) | -0.6 (0.73)
  CO2, Day 7: number analyzed (Participants) | 9 | 9
  CO2, Day 7 | 0.2 (1.48) | 0.3 (1.41)
  Chloride, Day 2: number analyzed (Participants) | 16 | 18
  Chloride, Day 2 | 0.3 (1.85) | -0.4 (1.89)
  Chloride, Day 5: number analyzed (Participants) | 8 | 9
  Chloride, Day 5 | 0.4 (2.00) | -0.9 (1.90)
  Chloride, Day 7: number analyzed (Participants) | 9 | 9
  Chloride, Day 7 | 0.4 (1.88) | 0.2 (2.33)
  Glucose, Day 2: number analyzed (Participants) | 16 | 18
  Glucose, Day 2 | -0.084 (0.1480) | 0.077 (0.2392)
  Glucose, Day 5: number analyzed (Participants) | 8 | 9
  Glucose, Day 5 | -0.160 (0.2754) | -0.256 (0.3867)
  Glucose, Day 7: number analyzed (Participants) | 9 | 9
  Glucose, Day 7 | 0.019 (0.3691) | -0.087 (0.2601)
  Potassium, Day 2: number analyzed (Participants) | 16 | 18
  Potassium, Day 2 | 0.01 (0.247) | 0.09 (0.289)
  Potassium, Day 5: number analyzed (Participants) | 8 | 9
  Potassium, Day 5 | -0.01 (0.476) | -0.08 (0.192)
  Potassium, Day 7: number analyzed (Participants) | 9 | 9
  Potassium, Day 7 | 0.01 (0.145) | 0.18 (0.393)
  Sodium, Day 2: number analyzed (Participants) | 16 | 18
  Sodium, Day 2 | -0.4 (1.41) | -0.3 (2.24)
  Sodium, Day 5: number analyzed (Participants) | 8 | 9
  Sodium, Day 5 | -0.8 (1.49) | -0.8 (1.86)
  Sodium, Day 7: number analyzed (Participants) | 9 | 9
  Sodium, Day 7 | 0.6 (1.33) | 1.2 (2.22)
  Urea nitrogen, Day 2: number analyzed (Participants) | 16 | 18
  Urea nitrogen, Day 2 | 0.228 (0.4467) | 0.628 (0.7585)
  Urea nitrogen, Day 5: number analyzed (Participants) | 8 | 9
  Urea nitrogen, Day 5 | -0.138 (0.6950) | 0.067 (0.8951)
  Urea nitrogen, Day 7: number analyzed (Participants) | 9 | 9
  Urea nitrogen, Day 7 | 0.321 (0.7415) | 0.441 (0.7504)
  Phosphate, Day 2: number analyzed (Participants) | 16 | 18
  Phosphate, Day 2 | 0.041 (0.0842) | 0.044 (0.0902)
  Phosphate, Day 5: number analyzed (Participants) | 8 | 9
  Phosphate, Day 5 | 0.014 (0.0983) | 0.012 (0.0349)
  Phosphate, Day 7: number analyzed (Participants) | 9 | 9
  Phosphate, Day 7 | 0.023 (0.0854) | 0.019 (0.0862)
  Triglycerides, Day 2: number analyzed (Participants) | 16 | 18
  Triglycerides, Day 2 | -0.111 (0.3084) | -0.121 (0.2674)
  Triglycerides, Day 5: number analyzed (Participants) | 8 | 9
  Triglycerides, Day 5 | -0.215 (0.3208) | -0.156 (0.2584)
  Triglycerides, Day 7: number analyzed (Participants) | 9 | 9
  Triglycerides, Day 7 | -0.089 (0.4124) | -0.031 (0.2996)
  Cholesterol, Day 2: number analyzed (Participants) | 16 | 18
  Cholesterol, Day 2 | 0.121 (0.4047) | 0.076 (0.2377)
  Cholesterol, Day 5: number analyzed (Participants) | 8 | 9
  Cholesterol, Day 5 | -0.036 (0.3000) | 0.113 (0.4685)
  Cholesterol, Day 7: number analyzed (Participants) | 9 | 9
  Cholesterol, Day 7 | -0.170 (0.4438) | -0.119 (0.4662)
  Anion gap, Day 2: number analyzed (Participants) | 16 | 18
  Anion gap, Day 2 | 0.5 (0.82) | 1.3 (0.96)
  Anion gap, Day 5: number analyzed (Participants) | 8 | 9
  Anion gap, Day 5 | 0.0 (1.41) | -0.3 (3.08)
  Anion gap, Day 7: number analyzed (Participants) | 9 | 9
  Anion gap, Day 7 | -0.1 (0.78) | 0.6 (1.42)

53. Secondary Outcome: Part 1: Change From Baseline in Clinical Chemistry Parameters: Lipase and Amylase
Description: Blood samples were collected to analyze the chemistry parameters: lipase and amylase. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Days 2, 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per Liter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Units per Liter
  Lipase, Day 2 | -0.4 (5.21) | 5.8 (13.57) | 3.2 (10.59)
  Lipase, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Lipase, Day 5 | 3.3 (3.33) | 1.3 (3.98) | 2.0 (9.92)
  Lipase, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Lipase, Day 7 | 4.5 (15.61) | -3.6 (19.59) | 2.1 (5.49)
  Amylase, Day 2 | 4.0 (5.54) | 3.9 (5.21) | 3.3 (8.70)
  Amylase, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Amylase, Day 5 | 5.5 (4.23) | 0.5 (4.32) | -1.2 (7.94)
  Amylase, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Amylase, Day 7 | 5.0 (9.08) | -0.7 (10.27) | 3.5 (9.23)

54. Secondary Outcome: Part 2: Change From Baseline in Clinical Chemistry Parameters: Lipase and Amylase
Description: as for outcome 53
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per Liter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Units per Liter
  Lipase, Day 2: number analyzed (Participants) | 16 | 18
  Lipase, Day 2 | -1.6 (5.77) | 0.3 (3.51)
  Lipase, Day 5: number analyzed (Participants) | 8 | 9
  Lipase, Day 5 | 2.3 (20.10) | 5.3 (13.17)
  Lipase, Day 7: number analyzed (Participants) | 9 | 9
  Lipase, Day 7 | -2.2 (8.77) | -0.1 (4.65)
  Amylase, Day 2: number analyzed (Participants) | 16 | 18
  Amylase, Day 2 | 0.8 (4.11) | 2.1 (3.83)
  Amylase, Day 5: number analyzed (Participants) | 8 | 9
  Amylase, Day 5 | 0.8 (7.42) | -0.7 (6.84)
  Amylase, Day 7: number analyzed (Participants) | 9 | 9
  Amylase, Day 7 | -0.3 (6.28) | 1.6 (4.39)

55. Secondary Outcome: Part 1: Change From Baseline in Clinical Chemistry Parameters: Albumin, Globulin and Protein
Description: Blood samples were collected to analyze the chemistry parameters: albumin, globulin and protein. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Days 2, 5, 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Grams per liter
  Albumin, Day 2 | 0.8 (2.65) | 0.7 (2.08) | 0.7 (1.49)
  Albumin, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Albumin, Day 5 | -0.8 (1.72) | 0.2 (2.32) | -0.2 (2.32)
  Albumin, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Albumin, Day 7 | 0.2 (2.14) | 0.0 (2.68) | 1.3 (1.49)
  Globulin, Day 2 | 1.0 (2.44) | 0.4 (1.80) | 1.2 (2.23)
  Globulin, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Globulin, Day 5 | 0.2 (2.40) | 0.2 (1.17) | 1.0 (2.10)
  Globulin, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Globulin, Day 7 | 0.0 (1.67) | -0.5 (2.33) | 0.6 (1.84)
  Protein, Day 2 | 1.8 (4.69) | 1.1 (3.65) | 1.9 (3.54)
  Protein, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Protein, Day 5 | -0.7 (2.80) | 0.3 (2.58) | 0.8 (3.13)
  Protein, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Protein, Day 7 | 0.2 (3.49) | -0.5 (4.56) | 1.9 (2.81)

56. Secondary Outcome: Part 2: Change From Baseline in Clinical Chemistry Parameters: Albumin, Globulin and Protein
Description: as for outcome 55
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 16 | 18
Grams per liter
  Albumin, Day 2 | 0.6 (2.78) | 0.2 (2.18)
  Albumin, Day 5: number analyzed (Participants) | 8 | 9
  Albumin, Day 5 | 0.9 (3.00) | 1.6 (4.36)
  Albumin, Day 7: number analyzed (Participants) | 9 | 9
  Albumin, Day 7 | 0.9 (2.47) | 0.4 (3.17)
  Globulin, Day 2 | 0.3 (1.98) | 0.8 (2.28)
  Globulin, Day 5: number analyzed (Participants) | 8 | 9
  Globulin, Day 5 | 0.8 (1.67) | 2.0 (2.78)
  Globulin, Day 7: number analyzed (Participants) | 9 | 9
  Globulin, Day 7 | -1.0 (3.08) | -0.1 (2.42)
  Protein, Day 2 | 0.9 (3.95) | 1.0 (3.33)
  Protein, Day 5: number analyzed (Participants) | 8 | 9
  Protein, Day 5 | 1.6 (3.85) | 3.6 (6.27)
  Protein, Day 7: number analyzed (Participants) | 9 | 9
  Protein, Day 7 | -0.1 (4.04) | 0.3 (4.58)

57. Secondary Outcome: Part 1: Change From Baseline in Clinical Chemistry Parameters: Creatinine, Direct Bilirubin, Bilirubin, and Urate
Description: Blood samples were collected to analyze the chemistry parameters: creatinine, direct bilirubin, bilirubin, and urate. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Days 2, 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Micromoles per liter
  Creatinine, Day 2 | 8.31 (4.422) | 7.12 (5.636) | 6.15 (4.228)
  Creatinine, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Creatinine, Day 5 | 3.10 (2.440) | 3.38 (3.026) | 1.92 (2.671)
  Creatinine, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Creatinine, Day 7 | 2.18 (5.799) | 0.97 (5.027) | 1.34 (6.215)
  Direct bilirubin, Day 2 | -0.12 (0.267) | -0.06 (0.329) | -0.01 (0.324)
  Direct bilirubin, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Direct bilirubin, Day 5 | -0.20 (0.261) | 0.02 (0.354) | 0.35 (0.138)
  Direct bilirubin, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Direct bilirubin, Day 7 | -0.03 (0.390) | -0.11 (0.330) | -0.11 (0.502)
  Bilirubin, Day 2 | -0.68 (1.327) | -0.39 (1.742) | -0.21 (1.236)
  Bilirubin, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Bilirubin, Day 5 | -1.85 (1.958) | -1.12 (1.306) | 0.55 (0.602)
  Bilirubin, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Bilirubin, Day 7 | 0.10 (1.638) | -1.06 (1.340) | -1.40 (2.078)
  Urate, Day 2 | -7.0 (17.31) | -7.9 (15.31) | -4.2 (21.77)
  Urate, Day 5: number analyzed (Participants) | 6 | 6 | 6
  Urate, Day 5 | -11.7 (8.36) | -7.0 (17.15) | 6.7 (30.59)
  Urate, Day 7: number analyzed (Participants) | 11 | 13 | 10
  Urate, Day 7 | -6.4 (28.61) | -6.8 (13.36) | 2.3 (20.74)

58. Secondary Outcome: Part 2: Change From Baseline in Clinical Chemistry Parameters: Creatinine, Direct Bilirubin, Bilirubin, and Urate
Description: as for outcome 57
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 16 | 18
Micromoles per liter
  Creatinine, Day 2 | 7.73 (4.766) | 6.97 (5.419)
  Creatinine, Day 5: number analyzed (Participants) | 8 | 9
  Creatinine, Day 5 | 3.54 (6.065) | 1.28 (6.361)
  Creatinine, Day 7: number analyzed (Participants) | 9 | 9
  Creatinine, Day 7 | 2.16 (3.830) | -0.98 (3.061)
  Direct bilirubin, Day 2 | 0.07 (0.328) | 0.04 (0.405)
  Direct bilirubin, Day 5: number analyzed (Participants) | 8 | 9
  Direct bilirubin, Day 5 | 0.13 (0.212) | 0.37 (0.374)
  Direct bilirubin, Day 7: number analyzed (Participants) | 9 | 9
  Direct bilirubin, Day 7 | -0.04 (0.300) | -0.12 (0.307)
  Bilirubin, Day 2 | 0.02 (1.518) | 0.31 (1.101)
  Bilirubin, Day 5: number analyzed (Participants) | 8 | 9
  Bilirubin, Day 5 | -0.41 (1.635) | 1.93 (2.272)
  Bilirubin, Day 7: number analyzed (Participants) | 9 | 9
  Bilirubin, Day 7 | -0.78 (2.499) | -0.08 (1.358)
  Urate, Day 2 | -12.4 (19.25) | 2.6 (15.74)
  Urate, Day 5: number analyzed (Participants) | 8 | 9
  Urate, Day 5 | -5.9 (12.97) | -2.0 (13.42)
  Urate, Day 7: number analyzed (Participants) | 9 | 9
  Urate, Day 7 | -6.0 (19.21) | -18.0 (22.32)

59. Secondary Outcome: Part 1: Absolute Values for Urinalysis Parameter: Specific Gravity
Description: Urine samples were collected to analyze the urinalysis parameter: specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1) and Days 2, 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Ratio
  Baseline (Day -1) | 1.0138 (0.00654) | 1.0168 (0.00685) | 1.0153 (0.00693)
  Day 2 | 1.0137 (0.00683) | 1.0150 (0.00766) | 1.0151 (0.00763)
  Day 5: number analyzed (Participants) | 6 | 6 | 6
  Day 5 | 1.0143 (0.00543) | 1.0197 (0.00638) | 1.0197 (0.00799)
  Day 7: number analyzed (Participants) | 11 | 13 | 10
  Day 7 | 1.0202 (0.00569) | 1.0159 (0.00760) | 1.0160 (0.00733)

60. Secondary Outcome: Part 2 : Absolute Values for Urinalysis Parameter: Specific Gravity
Description: as for outcome 59
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Ratio
  Baseline (Day -1) | 1.0146 (0.00742) | 1.0164 (0.00834)
  Day 2 | 1.0157 (0.00778) | 1.0182 (0.00906)
  Day 5: number analyzed (Participants) | 8 | 9
  Day 5 | 1.0123 (0.00715) | 1.0142 (0.01284)
  Day 7: number analyzed (Participants) | 9 | 9
  Day 7 | 1.0161 (0.01129) | 1.0144 (0.00735)

61. Secondary Outcome: Part 1: Absolute Values for Urinalysis Parameters: Potential of Hydrogen (pH)
Description: Urine samples were collected to analyze the urinalysis parameter: pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1) and Days 2, 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
pH
  Baseline (Day -1) | 6.18 (0.733) | 5.95 (0.631) | 5.88 (0.582)
  Day 2 | 6.16 (0.585) | 6.12 (0.723) | 6.20 (0.785)
  Day 5: number analyzed (Participants) | 6 | 6 | 6
  Day 5 | 5.83 (0.408) | 5.83 (0.258) | 5.75 (0.274)
  Day 7: number analyzed (Participants) | 11 | 13 | 10
  Day 7 | 5.82 (0.603) | 5.81 (0.596) | 6.15 (0.914)

62. Secondary Outcome: Part 1: Absolute Values for Urinalysis Parameter: Potential of Hydrogen
Description: as for outcome 61
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
pH
  Baseline (Day -1) | 6.12 (0.574) | 6.08 (0.354)
  Day 2 | 6.12 (0.452) | 6.17 (0.454)
  Day 5: number analyzed (Participants) | 8 | 9
  Day 5 | 6.13 (0.518) | 6.28 (0.565)
  Day 7: number analyzed (Participants) | 9 | 9
  Day 7 | 6.17 (0.433) | 5.94 (0.464)

63. Secondary Outcome: Part 1: Number of Participants With Urinalysis Dipstick Results: Glucose
Description: Urine samples were collected at indicated time points to analyze parameters including glucose by dipstick. Urinalysis included dipstick urine test which was used to screen for glucose. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters of urine glucose can be read as negative in the urine sample. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1) and Days 2, 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Participants
  Baseline (Day -1), Negative | 22 | 21 | 20
  Day 2, Negative | 22 | 21 | 20
  Day 5, Negative: number analyzed (Participants) | 6 | 6 | 6
  Day 5, Negative | 6 | 6 | 6
  Day 7, Negative: number analyzed (Participants) | 11 | 13 | 10
  Day 7, Negative | 11 | 13 | 10

64. Secondary Outcome: Part 2: Number of Participants With Urinalysis Dipstick Results: Glucose
Description: as for outcome 63
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Participants
  Baseline (Day -1), Negative | 17 | 18
  Day 2, Negative | 17 | 18
  Day 5, Negative: number analyzed (Participants) | 8 | 9
  Day 5, Negative | 8 | 9
  Day 7, Negative: number analyzed (Participants) | 9 | 9
  Day 7, Negative | 9 | 9

65. Secondary Outcome: Part 1: Number of Participants With Urinalysis Dipstick Results: Protein
Description: Urine samples were collected at indicated time points to analyze parameters including protein by dipstick. Urinalysis included dipstick urine test which was used to screen for protein. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters of urine protein can be read as negative, and trace in the urine sample. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1) and Days 2, 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Participants
  Baseline (Day -1), Negative | 22 | 21 | 20
  Day 2, Negative | 22 | 21 | 20
  Day 5, Negative: number analyzed (Participants) | 6 | 6 | 6
  Day 5, Negative | 6 | 6 | 6
  Day 7, Negative: number analyzed (Participants) | 11 | 13 | 10
  Day 7, Negative | 10 | 13 | 10
  Day 7, Trace: number analyzed (Participants) | 11 | 13 | 10
  Day 7, Trace | 1 | 0 | 0

66. Secondary Outcome: Part 2: Number of Participants With Urinalysis Dipstick Results: Protein
Description: as for outcome 65
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Participants
  Baseline (Day -1), Negative | 17 | 18
  Day 2, Negative | 17 | 18
  Day 5, Negative: number analyzed (Participants) | 8 | 9
  Day 5, Negative | 8 | 9
  Day 7, Negative: number analyzed (Participants) | 9 | 9
  Day 7, Negative | 8 | 9
  Day 7, Trace: number analyzed (Participants) | 9 | 9
  Day 7, Trace | 1 | 0

67. Secondary Outcome: Part 1: Number of Participants With Urinalysis Dipstick Results: Occult Blood
Description: Urine samples were collected at indicated time points to analyze parameters including occult blood by dipstick. Urinalysis included dipstick urine test which was used to screen for occult blood. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters of urine occult blood can be read as negative, trace, 1+, 2+, 3+ indicating proportional concentrations in the urine sample. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1) and Days 2, 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Participants
  Baseline (Day -1), Negative | 20 | 18 | 18
  Baseline (Day -1), Trace | 1 | 2 | 2
  Baseline (Day -1), 2+ | 1 | 1 | 0
  Day 2, Negative | 19 | 17 | 18
  Day 2, Trace | 2 | 3 | 1
  Day 2, 1+ | 0 | 0 | 1
  Day 2, 2+ | 1 | 0 | 0
  Day 2, 3+ | 0 | 1 | 0
  Day 5, Negative: number analyzed (Participants) | 6 | 6 | 6
  Day 5, Negative | 4 | 5 | 6
  Day 5, 1+: number analyzed (Participants) | 6 | 6 | 6
  Day 5, 1+ | 1 | 1 | 0
  Day 5, 2+: number analyzed (Participants) | 6 | 6 | 6
  Day 5, 2+ | 1 | 0 | 0
  Day 7, Negative: number analyzed (Participants) | 11 | 13 | 10
  Day 7, Negative | 10 | 11 | 9
  Day 7, Trace: number analyzed (Participants) | 11 | 13 | 10
  Day 7, Trace | 1 | 2 | 1

68. Secondary Outcome: Part 2: Number of Participants With Urinalysis Dipstick Results: Occult Blood
Description: as for outcome 67
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Participants
  Baseline (Day -1), Negative | 15 | 16
  Baseline (Day -1), Trace | 1 | 0
  Baseline (Day -1), 1+ | 0 | 1
  Baseline (Day -1), 2+ | 1 | 1
  Day 2, Negative | 17 | 17
  Day 2, 1+ | 0 | 1
  Day 5, Negative: number analyzed (Participants) | 8 | 9
  Day 5, Negative | 8 | 8
  Day 5, Trace: number analyzed (Participants) | 8 | 9
  Day 5, Trace | 0 | 1
  Day 7, Negative: number analyzed (Participants) | 9 | 9
  Day 7, Negative | 7 | 9
  Day 7, 1+: number analyzed (Participants) | 9 | 9
  Day 7, 1+ | 1 | 0
  Day 7, 2+: number analyzed (Participants) | 9 | 9
  Day 7, 2+ | 1 | 0

69. Secondary Outcome: Part 1: Number of Participants With Urinalysis Dipstick Results: Ketones
Description: Urine samples were collected at indicated time points to analyze parameters including ketones by dipstick. Urinalysis included dipstick urine test which was used to screen for ketones. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters of urine ketones can be read as negative, trace, 2+ indicating proportional concentrations in the urine sample. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1) and Days 2, 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Participants
  Baseline (Day -1), Negative | 22 | 20 | 20
  Baseline (Day -1), Trace | 0 | 1 | 0
  Day 2, Negative | 21 | 21 | 19
  Day 2, Trace | 1 | 0 | 1
  Day 5, Negative: number analyzed (Participants) | 6 | 6 | 6
  Day 5, Negative | 6 | 6 | 5
  Day 5, 2+: number analyzed (Participants) | 6 | 6 | 6
  Day 5, 2+ | 0 | 0 | 1
  Day 7, Negative: number analyzed (Participants) | 11 | 13 | 10
  Day 7, Negative | 10 | 13 | 10
  Day 7, Trace: number analyzed (Participants) | 11 | 13 | 10
  Day 7, Trace | 1 | 0 | 0

70. Secondary Outcome: Part 2: Number of Participants With Urinalysis Dipstick Results: Ketones
Description: Urine samples were collected at indicated time points to analyze parameters including ketones by dipstick. Urinalysis included dipstick urine test which was used to screen for ketones. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters of urine ketones can be read as negative, trace, 1+, 2+ indicating proportional concentrations in the urine sample. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Participants
  Baseline (Day -1), Negative | 17 | 17
  Baseline (Day -1), Trace | 0 | 1
  Day 2, Negative | 17 | 17
  Day 2, 1+ | 0 | 1
  Day 5, Negative: number analyzed (Participants) | 8 | 9
  Day 5, Negative | 8 | 7
  Day 5, Trace: number analyzed (Participants) | 8 | 9
  Day 5, Trace | 0 | 1
  Day 5, 2+: number analyzed (Participants) | 8 | 9
  Day 5, 2+ | 0 | 1
  Day 7, Negative: number analyzed (Participants) | 9 | 9
  Day 7, Negative | 8 | 9
  Day 7, Trace: number analyzed (Participants) | 9 | 9
  Day 7, Trace | 1 | 0

71. Secondary Outcome: Part 1: Number of Participants With Urinalysis Dipstick Results: Bilirubin and Nitrite
Description: Urine samples were collected at indicated time points to analyze parameters including bilirubin and nitrite by dipstick. Urinalysis included dipstick urine test which was used to screen for bilirubin and nitrite. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters of urine bilirubin and nitrite can be read as negative in the urine sample. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1) and Days 2, 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Participants
  Bilirubin, Baseline (Day -1), Negative | 22 | 21 | 20
  Bilirubin, Day 2, Negative | 22 | 21 | 20
  Bilirubin, Day 5, Negative: number analyzed (Participants) | 6 | 6 | 6
  Bilirubin, Day 5, Negative | 6 | 6 | 6
  Bilirubin, Day 7, Negative: number analyzed (Participants) | 11 | 13 | 10
  Bilirubin, Day 7, Negative | 11 | 13 | 10
  Nitrite, Baseline (Day -1), Negative | 22 | 21 | 20
  Nitrite, Day 2, Negative | 22 | 21 | 20
  Nitrite, Day 5, Negative: number analyzed (Participants) | 6 | 6 | 6
  Nitrite, Day 5, Negative | 6 | 6 | 6
  Nitrite, Day 7, Negative: number analyzed (Participants) | 11 | 13 | 10
  Nitrite, Day 7, Negative | 11 | 13 | 10

72. Secondary Outcome: Part 2: Number of Participants With Urinalysis Dipstick Results: Bilirubin and Nitrite
Description: as for outcome 71
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Participants
  Bilirubin, Baseline (Day -1), Negative | 17 | 18
  Bilirubin, Day 2, Negative | 17 | 18
  Bilirubin, Day 5, Negative: number analyzed (Participants) | 8 | 9
  Bilirubin, Day 5, Negative | 8 | 9
  Bilirubin, Day 7, Negative: number analyzed (Participants) | 9 | 9
  Bilirubin, Day 7, Negative | 9 | 9
  Nitrite, Baseline (Day -1), Negative | 17 | 18
  Nitrite, Day 2, Negative | 17 | 18
  Nitrite, Day 5, Negative: number analyzed (Participants) | 8 | 9
  Nitrite, Day 5, Negative | 8 | 9
  Nitrite, Day 7, Negative: number analyzed (Participants) | 9 | 9
  Nitrite, Day 7, Negative | 9 | 9

73. Secondary Outcome: Part 1: Number of Participants With Urinalysis Dipstick Results: Leukocyte Esterase
Description: Urine samples were collected at indicated time points to analyze parameters including leukocyte esterase by dipstick. Urinalysis included dipstick urine test which was used to screen for leukocyte esterase. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters of urine leukocyte esterase can be read as negative, trace, 1+ indicating proportional concentrations in the urine sample. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1) and Days 2, 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Participants
  Baseline (Day -1), Negative | 21 | 19 | 20
  Baseline (Day -1), Trace | 1 | 2 | 0
  Day 2, Negative | 22 | 19 | 20
  Day 2, 1+ | 0 | 2 | 0
  Day 5, Negative: number analyzed (Participants) | 6 | 6 | 6
  Day 5, Negative | 6 | 6 | 5
  Day 5, 1+: number analyzed (Participants) | 6 | 6 | 6
  Day 5, 1+ | 0 | 0 | 1
  Day 7, Negative: number analyzed (Participants) | 11 | 13 | 10
  Day 7, Negative | 9 | 12 | 10
  Day 7, Trace: number analyzed (Participants) | 11 | 13 | 10
  Day 7, Trace | 2 | 0 | 0
  Day 7, 1+: number analyzed (Participants) | 11 | 13 | 10
  Day 7, 1+ | 0 | 1 | 0

74. Secondary Outcome: Part 2: Number of Participants With Urinalysis Dipstick Results: Leukocyte Esterase
Description: Urine samples were collected at indicated time points to analyze parameters including leukocyte esterase by dipstick. Urinalysis included dipstick urine test which was used to screen for leukocyte esterase. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters of urine leukocyte esterase can be read as negative, trace indicating proportional concentrations in the urine sample. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period.
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Participants
  Baseline (Day -1), Negative | 17 | 17
  Baseline (Day -1), Trace | 0 | 1
  Day 2, Negative | 15 | 17
  Day 2, Trace | 2 | 1
  Day 5, Negative: number analyzed (Participants) | 8 | 9
  Day 5, Negative | 8 | 9
  Day 7, Negative: number analyzed (Participants) | 9 | 9
  Day 7, Negative | 9 | 9

75. Secondary Outcome: Part 1: Change From Baseline in Urinalysis Parameter: Specific Gravity
Description: Urine samples were collected to analyze the urinalysis parameter: specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Days 2, 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Ratio
  Day 2 | 0.0000 (0.00662) | -0.0017 (0.00770) | -0.0002 (0.00738)
  Day 5: number analyzed (Participants) | 6 | 6 | 6
  Day 5 | 0.0033 (0.00505) | 0.0043 (0.00524) | 0.0030 (0.00329)
  Day 7: number analyzed (Participants) | 11 | 13 | 10
  Day 7 | 0.0056 (0.00877) | -0.0014 (0.00957) | 0.0010 (0.00794)

76. Secondary Outcome: Part 2: Change From Baseline in Urinalysis Parameter: Specific Gravity
Description: as for outcome 75
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Ratio
  Day 2 | 0.0011 (0.00679) | 0.0018 (0.00899)
  Day 5: number analyzed (Participants) | 8 | 9
  Day 5 | -0.0005 (0.00447) | -0.0019 (0.01156)
  Day 7: number analyzed (Participants) | 9 | 9
  Day 7 | -0.0001 (0.00551) | -0.0022 (0.00748)

77. Secondary Outcome: Part 1: Change From Baseline for Urinalysis Parameter: Potential of Hydrogen
Description: Urine samples were collected to analyze the urinalysis parameter: pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visit, prior to the first study drug administration in each treatment period. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Days 2, 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
pH
  Day 2 | -0.02 (0.545) | 0.17 (0.796) | 0.33 (0.520)
  Day 5: number analyzed (Participants) | 6 | 6 | 6
  Day 5 | -0.58 (0.665) | -0.08 (0.585) | -0.08 (0.204)
  Day 7: number analyzed (Participants) | 11 | 13 | 10
  Day 7 | -0.45 (0.416) | -0.31 (0.723) | 0.15 (0.412)

78. Secondary Outcome: Part 2: Change From Baseline for Urinalysis Parameter: Potential of Hydrogen
Description: Urine samples were collected to analyze the urinalysis parameter: pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Days 2, 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
pH
  Day 2 | 0.00 (0.586) | 0.08 (0.393)
  Day 5: number analyzed (Participants) | 8 | 9
  Day 5 | 0.13 (0.354) | 0.11 (0.333)
  Day 7: number analyzed (Participants) | 9 | 9
  Day 7 | -0.06 (0.464) | -0.06 (0.635)

79. Secondary Outcome: Part 1: Number of Participants With Worst Case Urine Parameter: Glucose Results by Maximum Grade Increase Post-Baseline Relative to Baseline
Description: Urine samples were collected to analyze the urine parameter: glucose. Urinalysis parameters were graded according to Division of Acquired Immune Deficiency Syndrome (DAIDS) grading for severity of laboratory toxicities and clinical adverse events, version 2.1. The grades were grade 1 (mild), 2 (moderate), 3 (severe) and 4 (potentially life-threatening). Baseline was defined as the last assessment before the first dose of the study treatment. Only those urine parameters with maximum post-Baseline grade increase (Grade 1 to Grade 4) have been presented.
Time Frame: Up to Day 17
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Participants
  Increase to Grade 1 | 0 | 0 | 0
  Increase to Grade 2 | 0 | 0 | 0
  Increase to Grade 3 | 0 | 0 | 0
  Increase to Grade 4 | 0 | 0 | 0

80. Secondary Outcome: Part 2: Number of Participants With Worst Case Urine Parameter: Glucose Results by Maximum Grade Increase Post-Baseline Relative to Baseline
Description: as for outcome 79
Time Frame: Up to Day 9
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Participants
  Increase to Grade 1 | 0 | 0
  Increase to Grade 2 | 0 | 0
  Increase to Grade 3 | 0 | 0
  Increase to Grade 4 | 0 | 0

81. Secondary Outcome: Part 1: Number of Participants With Worst Case Urine Parameter: Protein Results by Maximum Grade Increase Post-Baseline Relative to Baseline
Description: Urine samples were collected to analyze the urine parameter: protein. Urinalysis parameters were graded according to Division of Acquired Immune Deficiency Syndrome (DAIDS) grading for severity of laboratory toxicities and clinical adverse events, version 2.1. The grades were grade 1 (mild), 2 (moderate), 3 (severe) and 4 (potentially life-threatening). Baseline was defined as the last assessment before the first dose of the study treatment. Only those urine parameters with maximum post-Baseline grade increase (Grade 1 to Grade 4) have been presented.
Time Frame: Up to Day 17
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Participants
  Increase to Grade 1 | 0 | 0 | 0
  Increase to Grade 2 | 0 | 0 | 0
  Increase to Grade 3 | 0 | 0 | 0
  Increase to Grade 4 | 0 | 0 | 0

82. Secondary Outcome: Part 2: Number of Participants With Worst Case Urine Parameter: Protein Results by Maximum Grade Increase Post-Baseline Relative to Baseline
Description: as for outcome 81
Time Frame: Up to Day 9
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Participants
  Increase to Grade 1 | 0 | 0
  Increase to Grade 2 | 0 | 0
  Increase to Grade 3 | 0 | 0
  Increase to Grade 4 | 0 | 0

83. Secondary Outcome: Part 1: Number of Participants With Worst Case Urine Parameter: Erythrocytes Results by Maximum Grade Increase Post-Baseline Relative to Baseline
Description: Urine samples were collected to analyze the urine parameter: erythrocytes. Urinalysis parameters were graded according to Division of Acquired Immune Deficiency Syndrome (DAIDS) grading for severity of laboratory toxicities and clinical adverse events, version 2.1. The grades were grade 1 (mild), 2 (moderate), 3 (severe) and 4 (potentially life-threatening). Baseline was defined as the last assessment before the first dose of the study treatment. Only those urine parameters with maximum post-Baseline grade increase (Grade 1 to Grade 4) have been presented.
Time Frame: Up to Day 17
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 8 | 7 | 4
Participants
  Increase to Grade 1 | 1 | 0 | 0
  Increase to Grade 2 | 0 | 0 | 0
  Increase to Grade 3 | 0 | 0 | 0
  Increase to Grade 4 | 0 | 0 | 0

84. Secondary Outcome: Part 2: Number of Participants With Worst Case Urine Parameter: Erythrocytes Results by Maximum Grade Increase Post-Baseline Relative to Baseline
Description: as for outcome 83
Time Frame: Up to Day 9
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Participants
  Increase to Grade 1 | 0 | 0
  Increase to Grade 2 | 0 | 0
  Increase to Grade 3 | 0 | 0
  Increase to Grade 4 | 0 | 0

85. Secondary Outcome: Part 1: Absolute Values of Electrocardiogram (ECG) Parameters: PR Interval, QRS Duration, QT Interval and QT Interval Corrected by Fridericia's Formula (QTcF)
Description: Twelve lead ECGs were obtained to measure PR interval, QRS duration, QT interval, and QTcF interval . Twelve lead ECGs were performed with the participant in a supine position after a rest of at least 10 minutes. Baseline was defined as the average of the triplicate pre-dose assessments within each treatment
Time Frame: Baseline (Day 1, pre-dose), and Day 1: 2, 4, 6 hours, and Day 5
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Milliseconds
  PR Interval, Baseline (Day1 pre-dose) | 162.8 (17.39) | 162.8 (18.05) | 163.1 (16.90)
  PR Interval, Day 1, 2 hours | 159.0 (18.13) | 158.0 (17.16) | 157.7 (17.78)
  PR Interval, Day 1, 4 hours | 159.2 (17.50) | 160.0 (17.51) | 159.9 (15.79)
  PR Interval, Day 1, 6 hours | 160.4 (18.70) | 158.2 (18.10) | 160.1 (16.87)
  PR Interval, Day 5: number analyzed (Participants) | 6 | 6 | 6
  PR Interval, Day 5 | 162.2 (16.02) | 170.8 (12.42) | 159.8 (31.98)
  QRS Duration, Baseline (Day 1) | 92.0 (7.09) | 93.1 (7.83) | 93.4 (8.61)
  QRS Duration, Day 1, 2 hours | 91.3 (7.12) | 92.8 (9.11) | 92.8 (8.15)
  QRS Duration, Day 1, 4 hours | 90.0 (8.16) | 91.5 (8.18) | 91.7 (9.04)
  QRS Duration, Day 1, 6 hours | 91.0 (7.67) | 91.7 (8.87) | 93.2 (8.63)
  QRS Duration, Day 5: number analyzed (Participants) | 6 | 6 | 6
  QRS Duration, Day 5 | 92.3 (4.93) | 94.2 (6.24) | 94.8 (9.99)
  QT Interval, Baseline (Day 1) | 397.0 (26.26) | 393.1 (29.10) | 394.2 (24.66)
  QT Interval, Day 1, 2 hours | 381.1 (24.29) | 375.0 (24.49) | 375.6 (19.77)
  QT Interval, Day 1, 4 hours | 391.2 (26.27) | 385.0 (23.31) | 386.4 (21.34)
  QT Interval, Day 1, 6 hours | 387.8 (21.90) | 379.3 (23.66) | 382.2 (20.88)
  QT Interval, Day 5: number analyzed (Participants) | 6 | 6 | 6
  QT Interval, Day 5 | 389.5 (18.32) | 374.8 (29.13) | 400.5 (9.01)
  QTcF Interval, Baseline (Day 1) | 404.3 (17.15) | 400.7 (19.60) | 403.7 (14.85)
  QTcF Interval, Day 1, 2 hours | 397.5 (18.03) | 393.1 (19.20) | 397.0 (15.11)
  QTcF Interval, Day 1, 4 hours | 399.1 (19.40) | 396.5 (399.3) | 399.3 (17.85)
  QTcF Interval, Day 1, 6 hours | 401.8 (17.12) | 398.4 (19.80) | 399.0 (16.65)
  QTcF Interval, Day 5: number analyzed (Participants) | 6 | 6 | 6
  QTcF Interval, Day 5 | 396.5 (23.48) | 399.0 (17.93) | 395.7 (13.69)

86. Secondary Outcome: Part 2: Absolute Values of ECG Parameters: PR Interval, QRS Duration, QT Interval and QTcF
Description: Twelve lead ECGs were obtained to measure PR interval, QRS duration, QT interval, and QTcF interval. Twelve lead ECGs were performed with the participant in a supine position after a rest of at least 10 minutes. Baseline was defined as the average of the triplicate pre-dose assessments within each treatment.
Time Frame: Baseline (Day 1, pre-dose), and Day 1: 2, 4, 6 hours, and Days 5, 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Milliseconds
  PR Interval, Baseline (Day 1 pre-dose) | 168.8 (15.94) | 170.9 (14.96)
  PR Interval, Day 1, 2 hours | 160.6 (14.92) | 167.0 (14.71)
  PR Interval, Day 1, 4 hours | 162.6 (17.19) | 167.4 (13.84)
  PR Interval, Day 1, 6 hours | 162.2 (15.23) | 160.9 (14.18)
  PR Interval, Day 5: number analyzed (Participants) | 8 | 9
  PR Interval, Day 5 | 172.1 (19.92) | 164.1 (9.69)
  PR Interval, Day 7: number analyzed (Participants) | 9 | 9
  PR Interval, Day 7 | 167.1 (9.09) | 176.2 (18.97)
  QRS Duration, Baseline (Day 1) | 89.8 (7.17) | 89.1 (5.71)
  QRS Duration, Day 1, 2 hours | 88.8 (6.87) | 87.9 (5.56)
  QRS Duration, Day 1, 4 hours | 87.5 (6.74) | 89.3 (6.49)
  QRS Duration, Day 1, 6 hours | 87.5 (6.50) | 89.7 (7.11)
  QRS Duration, Day 5: number analyzed (Participants) | 8 | 9
  QRS Duration, Day 5 | 87.8 (4.03) | 89.2 (8.51)
  QRS Duration, Day 7: number analyzed (Participants) | 9 | 9
  QRS Duration, Day 7 | 89.9 (6.83) | 88.8 (3.15)
  QT Interval, Baseline (Day 1) | 382.8 (16.73) | 383.6 (18.49)
  QT Interval, Day 1, 2 hours | 367.0 (15.73) | 385.2 (18.67)
  QT Interval, Day 1, 4 hours | 373.4 (11.37) | 391.8 (16.57)
  QT Interval, Day 1, 6 hours | 372.9 (16.48) | 367.8 (15.07)
  QT Interval, Day 5: number analyzed (Participants) | 8 | 9
  QT Interval, Day 5 | 367.8 (13.94) | 385.2 (25.34)
  QT Interval, Day 7: number analyzed (Participants) | 9 | 9
  QT Interval, Day 7 | 382.6 (17.92) | 378.2 (14.66)
  QTcF Interval, Baseline (Day 1) | 393.3 (11.84) | 390.9 (13.13)
  QTcF Interval, Day 1, 2 hours | 387.2 (12.56) | 390.3 (16.98)
  QTcF Interval, Day 1, 4 hours | 388.8 (11.52) | 392.3 (14.99)
  QTcF Interval, Day 1, 6 hours | 389.4 (11.52) | 390.2 (13.13)
  QTcF Interval, Day 5: number analyzed (Participants) | 8 | 9
  QTcF Interval, Day 5 | 388.6 (7.63) | 395.3 (14.71)
  QTcF Interval, Day 7: number analyzed (Participants) | 9 | 9
  QTcF Interval, Day 7 | 395.3 (12.11) | 381.1 (9.78)

87. Secondary Outcome: Part 1: Change From Baseline in ECG Parameters: PR Interval, QRS Duration, QT Interval and QTcF Interval
Description: Twelve lead ECGs were obtained to measure PR interval, QRS duration, QT interval, QTcF interval. Twelve lead ECGs were performed with the participant in a supine position after a rest of at least 10 minutes. Baseline was defined as the average of the triplicate pre-dose assessments within each treatment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose), and Day 1: 2, 4, 6 hours, and Day 5
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Milliseconds
  PR Interval, Day 1, 2 hours | -3.8 (10.19) | -4.7 (7.79) | -5.5 (11.16)
  PR Interval, Day 1, 4 hours | -3.6 (10.28) | -2.8 (6.31) | -3.3 (9.04)
  PR Interval, Day 1, 6 hours | -2.5 (9.65) | -4.6 (11.29) | -3.0 (10.31)
  PR Interval, Day 5: number analyzed (Participants) | 6 | 6 | 6
  PR Interval, Day 5 | 2.8 (9.13) | -1.8 (8.28) | -6.0 (9.44)
  QRS Duration, Day 1, 2 hours | -0.7 (4.22) | -0.4 (4.60) | -0.7 (3.12)
  QRS Duration, Day 1, 4 hours | -2.0 (4.40) | -1.6 (5.00) | -1.7 (3.54)
  QRS Duration, Day 1, 6 hours | -1.0 (4.55) | -1.4 (3.99) | -0.3 (2.45)
  QRS Duration, Day 5: number analyzed (Participants) | 6 | 6 | 6
  QRS Duration, Day 5 | 2.0 (3.46) | -1.3 (4.97) | -0.8 (2.14)
  QT Interval, Day 1, 2 hours | -15.8 (11.54) | -18.1 (10.24) | -18.6 (11.71)
  QT Interval, Day 1, 4 hours | -5.8 (14.45) | -8.1 (13.18) | -7.9 (11.78)
  QT Interval, Day 1, 6 hours | -9.1 (12.89) | -13.8 (13.51) | -12.0 (13.81)
  QT Interval, Day 5: number analyzed (Participants) | 6 | 6 | 6
  QT Interval, Day 5 | 0.8 (14.27) | -14.8 (19.54) | -14.5 (9.85)
  QTcF Interval, Day 1, 2 hours | -6.8 (7.36) | -7.6 (6.58) | -6.8 (6.32)
  QTcF Interval, Day 1, 4 hours | -5.1 (9.07) | -4.2 (8.58) | -4.5 (6.88)
  QTcF Interval, Day 1, 6 hours | -2.5 (8.72) | -2.2 (9.87) | -4.7 (7.34)
  QTcF Interval, Day 5: number analyzed (Participants) | 6 | 6 | 6
  QTcF Interval, Day 5 | -6.0 (14.04) | -2.3 (14.31) | -5.8 (8.16)

88. Secondary Outcome: Part 2: Change From Baseline in ECG Parameters: PR Interval, QRS Duration, QT Interval and QTcF Interval
Description: as for outcome 87
Time Frame: Baseline (Day 1, pre-dose), and Day 1: 2, 4, 6 hours, Days 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Milliseconds
  PR Interval, Day 1, 2 hours | -8.1 (10.19) | -3.9 (8.27)
  PR Interval, Day 1, 4 hours | -6.1 (12.06) | -3.4 (9.73)
  PR Interval, Day 1, 6 hours | -6.5 (10.71) | -9.9 (12.21)
  PR Interval, Day 5: number analyzed (Participants) | 8 | 9
  PR Interval, Day 5 | -4.5 (10.94) | -4.8 (8.84)
  PR Interval, Day 7: number analyzed (Participants) | 9 | 9
  PR Interval, Day 7 | 5.3 (7.89) | 3.3 (11.88)
  QRS Duration, Day 1, 2 hours | -1.0 (5.14) | -1.2 (2.56)
  QRS Duration, Day 1, 4 hours | -2.3 (5.39) | 0.2 (2.21)
  QRS Duration Day 1, 6 hours | -2.2 (4.97) | 0.6 (2.75)
  QRS Duration, Day 5: number analyzed (Participants) | 8 | 9
  QRS Duration, Day 5 | -3.8 (7.74) | 0.0 (2.74)
  QRS Duration, Day 7: number analyzed (Participants) | 9 | 9
  QRS Duration, Day 7 | 1.7 (3.12) | -0.2 (3.93)
  QT Interval, Day 1, 2 hours | -15.8 (13.03) | 1.6 (11.34)
  QT Interval, Day 1, 4 hours | -9.5 (13.61) | 8.2 (10.80)
  QT Interval, Day 1, 6 hours | -9.9 (14.35) | -15.7 (10.87)
  QT Interval, Day 5: number analyzed (Participants) | 8 | 9
  QT Interval, Day 5 | -16.0 (17.47) | -2.3 (19.62)
  QT Interval, Day 7: number analyzed (Participants) | 9 | 9
  QT Interval, Day 7 | 0.6 (8.03) | -1.3 (16.72)
  QTcF Interval, Day 1, 2 hours | -6.1 (11.76) | -0.6 (8.47)
  QTcF Interval, Day 1, 4 hours | -4.5 (8.52) | 1.4 (7.88)
  QTcF Interval, Day 1, 6 hours | -3.9 (5.96) | -0.8 (8.05)
  QTcF Interval, Day 5: number analyzed (Participants) | 8 | 9
  QTcF Interval, Day 5 | -0.5 (6.26) | 0.2 (9.56)
  QTcF Interval, Day 7: number analyzed (Participants) | 9 | 9
  QTcF Interval, Day 7 | -1.7 (6.48) | -5.7 (11.38)

89. Secondary Outcome: Part 1: Absolute Values of Vital Sign Parameters: Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: SBP and DBP were measured in the semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline is defined as the average of the triplicate predose assessments within each treatment.
Time Frame: Baseline (Day 1, pre-dose), and Day 1: 24, 48, 72 hours, Days 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Millimeters of mercury
  DBP, Baseline (Day 1) | 61.5 (6.39) | 63.2 (7.21) | 63.2 (9.05)
  DBP, Day 1, 24 hours | 60.9 (7.34) | 63.1 (8.18) | 63.0 (6.40)
  DBP, Day 1, 48 hours: number analyzed (Participants) | 18 | 19 | 16
  DBP, Day 1, 48 hours | 59.8 (5.89) | 61.2 (6.68) | 59.6 (4.72)
  DBP, Day 1, 72 hours: number analyzed (Participants) | 6 | 6 | 6
  DBP, Day 1, 72 hours | 58.7 (6.19) | 63.0 (8.69) | 61.3 (4.08)
  DBP, Day 5: number analyzed (Participants) | 6 | 6 | 6
  DBP, Day 5 | 61.7 (5.24) | 64.2 (6.05) | 61.5 (4.18)
  DBP Interval, Day 7: number analyzed (Participants) | 11 | 13 | 10
  DBP Interval, Day 7 | 62.0 (8.46) | 61.0 (7.18) | 59.4 (5.48)
  SBP, Baseline (Day 1) | 108.9 (11.23) | 110.6 (13.47) | 110.8 (16.32)
  SBP, Day 1, 24 hours | 106.1 (10.41) | 112.9 (13.30) | 108.7 (10.54)
  SBP, Day 1, 48 hours: number analyzed (Participants) | 18 | 19 | 16
  SBP, Day 1, 48 hours | 104.7 (8.60) | 110.5 (14.02) | 106.7 (10.47)
  SBP, Day 1, 72 hours: number analyzed (Participants) | 6 | 6 | 6
  SBP, Day 1, 72 hours | 100.5 (6.53) | 114.7 (21.57) | 112.2 (12.19)
  SBP, Day 5: number analyzed (Participants) | 6 | 6 | 6
  SBP, Day 5 | 105.8 (8.64) | 118.0 (19.67) | 109.2 (10.98)
  SBP, Day 7: number analyzed (Participants) | 11 | 13 | 10
  SBP, Day 7 | 110.5 (13.40) | 108.2 (9.24) | 106.8 (11.94)

90. Secondary Outcome: Part 2: Absolute Values of Vital Signs: DBP and SBP
Description: SBP and DBP were measured in the semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the average of the triplicate predose assessments within each treatment.
Time Frame: Baseline (Day 1, pre-dose), and Day 1: 24, 48 hours, Days 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Millimeters of mercury
  DBP, Baseline (Day 1 pre-dose) | 65.1 (8.39) | 65.7 (9.26)
  DBP, Day 1, 24 hours | 64.0 (6.44) | 62.9 (9.09)
  DBP, Day 1, 48 hours | 61.8 (7.89) | 61.1 (9.78)
  DBP, Day 5: number analyzed (Participants) | 8 | 9
  DBP, Day 5 | 68.1 (4.49) | 60.0 (4.30)
  DBP Interval, Day 7: number analyzed (Participants) | 9 | 9
  DBP Interval, Day 7 | 62.2 (7.63) | 67.6 (7.60)
  SBP, Baseline (Day 1 pre-dose) | 110.9 (9.39) | 111.5 (11.73)
  SBP, Day 1, 24 hours | 110.1 (10.84) | 110.4 (13.49)
  SBP, Day 1, 48 hours | 108.4 (10.06) | 106.9 (9.58)
  SBP, Day 5: number analyzed (Participants) | 8 | 9
  SBP, Day 5 | 113.3 (5.97) | 108.7 (9.31)
  SBP, Day 7: number analyzed (Participants) | 9 | 9
  SBP, Day 7 | 105.8 (6.28) | 108.4 (9.30)

91. Secondary Outcome: Part 1: Absolute Values of Vital Signs: Pulse Rate
Description: Pulse rate was measured in the semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the average of the triplicate predose assessments within each treatment.
Time Frame: Baseline (Day 1, pre-dose), and Day 1: 24, 48, 72 hours, Days 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Beats per minute
  Baseline (Day 1, Pre-dose) | 64.9 (13.41) | 66.06 (14.53) | 67.4 (14.19)
  Day 1, 24 hours | 61.7 (9.05) | 68.6 (11.69) | 64.8 (11.47)
  Day 1, 48 hours: number analyzed (Participants) | 18 | 19 | 16
  Day 1, 48 hours | 61.7 (6.88) | 65.5 (11.81) | 64.9 (10.20)
  Day 1, 72 hours: number analyzed (Participants) | 6 | 6 | 6
  Day 1, 72 hours | 61.2 (10.76) | 77.7 (22.98) | 57.7 (10.76)
  Day 5: number analyzed (Participants) | 6 | 6 | 6
  Day 5 | 62.3 (6.06) | 77.5 (20.84) | 59.7 (11.81)
  Day 7: number analyzed (Participants) | 11 | 13 | 10
  Day 7 | 58.9 (8.29) | 60.8 (8.49) | 69.6 (9.83)

92. Secondary Outcome: Part 2: Absolute Values of Vital Signs: Pulse Rate
Description: as for outcome 91
Time Frame: Baseline (Day 1, pre-dose), and Day 1: 24, 48 hours, Day 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Beats per minute
  Baseline (Day 1, pre-dose) | 64.4 (5.76) | 64.2 (7.34)
  Day 1, 24 hours | 65.7 (9.22) | 67.3 (8.21)
  Day 1, 48 hours | 66.9 (7.29) | 69.1 (8.33)
  Day 5: number analyzed (Participants) | 8 | 9
  Day 5 | 70.0 (7.29) | 66.8 (7.10)
  Day 7: number analyzed (Participants) | 9 | 9
  Day 7 | 65.9 (5.64) | 62.2 (7.12)

93. Secondary Outcome: Part 1: Absolute Values of Vital Signs: Oral Temperature
Description: Oral temperature were measured in the semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the average of the triplicate predose assessments within each treatment.
Time Frame: Baseline (Day 1, pre-dose), and Day 1: 24, 48, 72 hours, Days 5, 6 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Degrees celsius
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Degrees celsius
  Baseline (Day 1 pre-dose) | 36.38 (0.424) | 36.43 (0.451) | 36.52 (0.382)
  Day 1, 24 hours | 36.47 (0.431) | 36.55 (0.481) | 36.60 (0.422)
  Day 1, 48 hours: number analyzed (Participants) | 18 | 19 | 16
  Day 1, 48 hours | 36.54 (0.343) | 36.54 (0.385) | 36.61 (0.264)
  Day 1, 72 hours: number analyzed (Participants) | 6 | 6 | 6
  Day 1, 72 hours | 36.45 (0.423) | 36.77 (0.314) | 36.25 (0.505)
  Day 5: number analyzed (Participants) | 18 | 19 | 16
  Day 5 | 36.44 (0.475) | 36.43 (0.527) | 36.48 (0.355)
  Day 6: number analyzed (Participants) | 12 | 13 | 10
  Day 6 | 36.43 (0.317) | 36.49 (0.468) | 36.43 (0.267)
  Day 7: number analyzed (Participants) | 11 | 13 | 10
  Day 7 | 36.51 (0.501) | 36.46 (0.380) | 36.72 (0.282)

94. Secondary Outcome: Part 2: Absolute Values of Vital Signs: Oral Temperature
Description: as for outcome 93
Time Frame: Baseline (Day 1, pre-dose), and Day 1: 24, 48 hours, Day 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Degree celsius
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Degree celsius
  Baseline (Day 1, pre-dose) | 36.28 (0.366) | 36.30 (0.230)
  Day 1, 24 hours | 36.42 (0.325) | 36.33 (0.307)
  Day 1, 48 hours | 36.42 (0.321) | 36.32 (0.349)
  Day 5: number analyzed (Participants) | 17 | 17
  Day 5 | 36.41 (0.347) | 36.31 (0.313)
  Day 6: number analyzed (Participants) | 9 | 9
  Day 6 | 36.43 (0.339) | 36.18 (0.377)
  Day 7: number analyzed (Participants) | 9 | 9
  Day 7 | 36.57 (0.269) | 36.38 (0.402)

95. Secondary Outcome: Part 1: Absolute Values of Vital Signs: Respiratory Rate
Description: Respiratory rate was measured in the semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the average of the triplicate predose assessments within each treatment.
Time Frame: Baseline (Day 1, pre-dose), and Day 1: 24, 48, 72 hours, Days 5 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Breaths per minute
  Baseline (Day 1, pre-dose) | 14.1 (2.65) | 13.6 (2.58) | 13.9 (3.28)
  Day 1, 24 hours | 13.8 (3.26) | 13.8 (3.03) | 14.8 (2.93)
  Day 1, 48 hours: number analyzed (Participants) | 18 | 19 | 16
  Day 1, 48 hours | 14.9 (2.68) | 12.7 (2.42) | 14.1 (2.00)
  Day 1, 72 hours: number analyzed (Participants) | 6 | 6 | 6
  Day 1, 72 hours | 14.0 (2.83) | 13.0 (2.45) | 14.0 (1.26)
  Day 5: number analyzed (Participants) | 6 | 6 | 6
  Day 5 | 11.7 (3.44) | 12.0 (2.83) | 14.7 (3.93)
  Day 7: number analyzed (Participants) | 11 | 13 | 10
  Day 7 | 14.0 (2.97) | 14.6 (1.89) | 12.9 (3.78)

96. Secondary Outcome: Part 2: Absolute Values of Vital Signs: Respiratory Rate
Description: as for outcome 95
Time Frame: Baseline (Day 1, pre-dose), and Day 1: 24, 48 hours, Days 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Breaths per minute
  Baseline (Day 1, pre-dose) | 12.7 (2.34) | 12.9 (2.49)
  Day 1, 24 hours | 14.5 (1.94) | 13.9 (2.52)
  Day 1, 48 hours | 13.1 (2.84) | 13.8 (2.37)
  Day 5: number analyzed (Participants) | 8 | 9
  Day 5 | 11.3 (2.38) | 12.4 (3.13)
  Day 7: number analyzed (Participants) | 9 | 9
  Day 7 | 13.5 (2.07) | 13.1 (1.45)

97. Secondary Outcome: Part 1: Change From Baseline in Vital Signs: DBP and SBP
Description: SBP and DBP were measured in the semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the average of the triplicate predose assessments within each treatment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, pre-dose), and Day 1: 24, 48, 72 hours, Days 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Millimeters of mercury
  DBP, Day 1, 24 hours | -0.6 (5.27) | -0.1 (7.40) | 13.9 (7.45)
  DBP, Day 1, 48 hours: number analyzed (Participants) | 18 | 19 | 16
  DBP, Day 1, 48 hours | -2.4 (5.21) | -2.5 (5.25) | -2.4 (5.66)
  DBP, Day 1, 72 hours: number analyzed (Participants) | 6 | 6 | 6
  DBP, Day 1, 72 hours | -4.2 (6.52) | -1.3 (6.86) | -1.5 (6.66)
  DBP, Day 5: number analyzed (Participants) | 6 | 6 | 6
  DBP, Day 5 | -1.2 (6.18) | -0.2 (7.25) | -1.3 (5.20)
  DBP, Day 7: number analyzed (Participants) | 11 | 13 | 10
  DBP, Day 7 | -0.1 (7.49) | -2.3 (5.76) | -2.1 (8.01)
  SBP, Day 1, 24 hours | -2.8 (9.63) | 2.3 (7.37) | -2.1 (9.95)
  SBP, Day 1, 48 hours: number analyzed (Participants) | 18 | 19 | 16
  SBP, Day 1, 48 hours | -4.0 (6.08) | -0.5 (6.57) | -3.8 (10.80)
  SBP, Day 1, 72 hours: number analyzed (Participants) | 6 | 6 | 6
  SBP, Day 1, 72 hours | -7.8 (9.09) | 2.8 (8.64) | 4.2 (6.74)
  SBP, Day 5: number analyzed (Participants) | 6 | 6 | 6
  SBP, Day 5 | -2.5 (7.06) | 6.2 (9.13) | 1.2 (6.52)
  SBP, Day 7: number analyzed (Participants) | 11 | 13 | 10
  SBP, Day 7 | 1.4 (7.63) | -2.4 (10.06) | -5.1 (10.71)

98. Secondary Outcome: Part 2: Change From Baseline in Vital Signs: DBP and SBP
Description: as for outcome 97
Time Frame: Baseline (Day 1, pre-dose), and Day 1: 24, 48 hours, Days 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Millimeters of mercury
  DBP, Day 1, 24 hours | -1.1 (4.34) | -2.8 (7.18)
  DBP, Day 1, 48 hours | -3.3 (6.30) | -4.6 (5.28)
  DBP, Day 5: number analyzed (Participants) | 8 | 9
  DBP, Day 5 | -0.3 (6.96) | -1.8 (5.54)
  DBP Interval, Day 7: number analyzed (Participants) | 9 | 9
  DBP Interval, Day 7 | 0.1 (4.48) | -2.0 (6.61)
  SBP, Day 1, 24 hours | -0.8 (9.19) | -1.1 (10.57)
  SBP, Day 1, 48 hours | -2.5 (5.56) | -4.6 (7.81)
  SBP, Day 5: number analyzed (Participants) | 8 | 9
  SBP, Day 5 | 1.3 (10.10) | 1.9 (8.22)
  SBP, Day 7: number analyzed (Participants) | 9 | 9
  SBP, Day 7 | -4.1 (4.48) | -7.8 (8.74)

99. Secondary Outcome: Part 1: Change From Baseline in Vital Signs: Pulse Rate
Description: Pulse rate was measured in the semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the average of the triplicate predose assessments within each treatment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, pre-dose), and Day 1: 24, 48, 72 hours, Days 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Beats per minute
  Day 1, 24 hours | -3.2 (8.87) | 2.6 (8.69) | -2.7 (10.80)
  Day 1, 48 hours: number analyzed (Participants) | 18 | 19 | 16
  Day 1, 48 hours | -0.7 (9.60) | -1.4 (8.38) | -2.8 (10.94)
  Day 1, 72 hours: number analyzed (Participants) | 6 | 6 | 6
  Day 1, 72 hours | -5.2 (14.32) | 7.2 (5.98) | 0.7 (4.41)
  Day 5: number analyzed (Participants) | 6 | 6 | 6
  Day 5 | -4.0 (9.08) | 7.0 (6.32) | 2.7 (5.89)
  Day 7: number analyzed (Participants) | 11 | 13 | 10
  Day 7 | -1.0 (7.33) | -4.4 (9.63) | -4.4 (9.42)

100. Secondary Outcome: Part 2: Change From Baseline in Vital Signs: Pulse Rate
Description: as for outcome 99
Time Frame: Baseline (Day 1, pre-dose), and Day 1: 24, 48 hours, Days 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Beats per minute
  Day 1, 24 hours | 1.3 (9.68) | 3.1 (8.32)
  Day 1, 48 hours | 2.5 (5.37) | 4.9 (8.36)
  Day 5: number analyzed (Participants) | 8 | 9
  Day 5 | 7.0 (8.19) | 3.4 (5.32)
  Day 7: number analyzed (Participants) | 9 | 9
  Day 7 | 0.2 (4.18) | -2.9 (6.51)

101. Secondary Outcome: Part 1: Change From Baseline in Vital Signs: Oral Temperature
Description: Oral temperature was measured in the semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the average of the triplicate predose assessments within each treatment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, pre-dose), and Day 1: 24, 48, 72 hours, Days 5, 6 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Degrees Celsius
  Day 1, 24 hours | 0.09 (0.507) | 0.11 (0.479) | 0.08 (0.443)
  Day 1, 48 hours: number analyzed (Participants) | 18 | 19 | 16
  Day 1, 48 hours | 0.15 (0.485) | 0.05 (0.415) | 0.11 (0.274)
  Day 1, 72 hours: number analyzed (Participants) | 6 | 6 | 6
  Day 1, 72 hours | -0.03 (0.497) | 0.38 (0.313) | -0.03 (0.314)
  Day 5: number analyzed (Participants) | 18 | 19 | 16
  Day 5 | 0.05 (0.418) | -0.06 (0.494) | -0.03 (0.401)
  Day 6: number analyzed (Participants) | 12 | 13 | 10
  Day 6 | 0.08 (0.541) | -0.04 (0.435) | -0.20 (0.521)
  Day 7: number analyzed (Participants) | 11 | 13 | 10
  Day 7 | 0.17 (0.443) | -0.07 (0.523) | 0.09 (0.300)

102. Secondary Outcome: Part 2: Change From Baseline in Vital Signs: Oral Temperature
Description: Oral temperature was measured in the semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, pre-dose), and Day 1: 24, 48 hours, Days 5, 6 and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Degrees Celsius
  Day 1, 24 hours | 0.14 (0.378) | 0.03 (0.341)
  Day 1, 48 hours | 0.14 (0.326) | 0.02 (0.350)
  Day 5: number analyzed (Participants) | 17 | 17
  Day 5 | 0.12 (0.385) | 0.01 (0.356)
  Day 6: number analyzed (Participants) | 9 | 9
  Day 6 | 0.11 (0.314) | -0.19 (0.481)
  Day 7: number analyzed (Participants) | 9 | 9
  Day 7 | 0.24 (0.167) | 0.01 (0.470)

103. Secondary Outcome: Part 1: Change From Baseline in Vital Signs: Respiratory Rate
Description: Respiratory rate was measured in the semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the average of the triplicate predose assessments within each treatment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, pre-dose), and Day 1: 24, 48 hours, Days 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet)
Number analyzed (Participants) | 22 | 21 | 20
Breaths per minute
  Day 1, 24 hours | -0.3 (2.57) | 0.2 (3.84) | 0.9 (2.86)
  Day 1, 48 hours: number analyzed (Participants) | 18 | 19 | 16
  Day 1, 48 hours | 0.9 (3.64) | -0.8 (3.67) | 0.5 (2.58)
  Day 1, 72 hours: number analyzed (Participants) | 6 | 6 | 6
  Day 1, 72 hours | -1.3 (2.07) | -1.3 (3.01) | -0.3 (2.34)
  Day 5: number analyzed (Participants) | 6 | 6 | 6
  Day 5 | -3.7 (2.94) | -2.3 (4.63) | 0.3 (3.44)
  Day 7: number analyzed (Participants) | 11 | 13 | 10
  Day 7 | 0.4 (4.37) | 1.4 (2.22) | -0.3 (3.40)

104. Secondary Outcome: Part 2: Change From Baseline in Vital Signs: Respiratory Rate
Description: as for outcome 103
Time Frame: Baseline (Day 1, pre-dose), and Day 1: 24, 48 hours, Days 5, and 7
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
Number analyzed (Participants) | 17 | 18
Breaths per minute
  Day 1, 24 hours | 1.8 (2.82) | 1.0 (3.01)
  Day 1, 48 hours | 0.4 (3.48) | 0.9 (3.01)
  Day 5: number analyzed (Participants) | 8 | 9
  Day 5 | -1.0 (3.02) | -1.3 (4.24)
  Day 7: number analyzed (Participants) | 8 | 9
  Day 7 | 0.0 (2.83) | 1.1 (3.33)

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to Day 17 in Part 1 and up to Day 9 in Part 2
Description: Safety Population consisted of all participants who received at least one dose of study intervention.
Arm/Group | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet) | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21 | 0/20 | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/20 | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 1/20 | 1/17 | 2/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1:Treatment A:GSK3640254 25mg+GSK3640254 100mg+DTG 50 mg (N=22) | Part 1:Treatment B:GSK3640254/DTG 150/50 mg(Monolayer Tablet) (N=21) | Part 1:Treatment C:GSK3640254/DTG 150/50mg(Bilayer Tablet) (N=20) | Part 2: Treatment D: GSK3640254/DTG, 150 mg/50 mg (Fed) (N=17) | Part 2: Treatment E: GSK3640254/DTG, 150 mg/50 mg (Fasted) (N=18)
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/92/NCT04857892/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT04857892/SAP_001.pdf